# Clinical Trial Protocol: THR-1442-C-480

**Study Title:** A Phase 3, Randomized, Double-Blind, Active-Controlled Study to

Evaluate the Effects of Bexagliflozin versus Glimepiride in Subjects with Type 2 Diabetes Mellitus Who Have Inadequate Glycemic

Control by Metformin

Study Number: THR-1442-C-480

**Study Phase:** 3

**Product Name:** Bexagliflozin Tablets **Indication:** Type 2 Diabetes Mellitus

**Investigators:** Multicenter study **EudraCT Number:** 2016-002013-21

**IND Number:** 103822

**Sponsor:** Theracos Sub, LLC

**Sponsor Contact:** Annie Conery, Ph.D.

Project Manager

Translational Medicine Group Massachusetts General Hospital

185 Cambridge Street, Boston, MA 02114

Phone: 1-617-726-5930 Fax: 617-643-8203

E-mail: aconery@mgh.harvard.edu

**Medical Monitor:** J. Paul Lock, M.D.

Theracos Sub, LLC

225 Cedar Hill Road, Suite 200, Marlborough, MA 01752

Phone: 1-508-735-9491 Fax: 617-643-8203

E-mail: jplock@theracos.com

| | Date |
|--------------|-----------------|
| Version 3.0: | 27 October 2016 |

### **Confidentiality Statement**

The information in this document is the confidential information of Theracos Sub, LLC ("Theracos") and must not be disclosed, used, or copied except with prior written approval from Theracos or to the extent required by applicable laws, rules and regulations.

# **TABLE OF CONTENTS**

| SY | NOPSIS | | 7 |
|---|---|---|---|
| LI | ST OF AB | BREVIATIONS AND DEFINITIONS OF TERMS | 13 |
| 1 | INTROI | DUCTION | 16 |
| | 1.1 Ty | pe 2 Diabetes Mellitus | 16 |
| | 1.2 Be | exagliflozin for the Treatment of Type 2 Diabetes Mellitus | 17 |
| 2 | STUDY | OBJECTIVES | 18 |
| | 2.1 Pr | imary Objective | 18 |
| | 2.2 Ke | ey Secondary Objectives | 18 |
| | 2.3 Ex | xploratory Objectives | 18 |
| 3 | INVEST | TIGATIONAL PLAN | 20 |
| | 3.1 O | verall Study Design and Plan | 20 |
| | 3.2 Ra | ationale for Study Design and Control Group | 20 |
| | 3.2.1 | Rationale for Background Medication and Active Comparator | 20 |
| | 3.2.2 | Rationale for the Study Design | 21 |
| | 3.2.3 | Rationale for the Dose Selection | 21 |
| | 3.3 Re | esearch Methods and Procedures | 22 |
| | 3.3.1 | Wash-out and Run-in Period | 22 |
| | 3.3.2 | Treatment Period | 23 |
| | 3 | 3.2.1 Glimepiride Dose Titration | 24 |
| | 3.3.3 | Glycemic Control Monitoring | |
| | | Wash-out Period and Placebo Run-in Period | |
| | | Treatment Period | |
| | 3.3.4 | Other Safety Monitoring Activities | |
| | 3.3.5 | Data and Safety Monitoring Board (DSMB) | |
| | 3.3.6 | Major Adverse Cardiovascular Event (MACE) Adjudication | |
| | 3.3.7 | Diabetic Ketoacidosis (DKA) Event Adjudication | |
| | | udy Duration and Dates | |
| 4 | | POPULATION SELECTION | |
| _ | | udy Population | |
| | | clusion Criteria | |
| | | clusion Criteria | |
| 5 | | TREATMENTS | |
| J | | escription of Treatments | |
| | 5.1.1 | Investigational Product | |
| | | Active Comparator | 32 |

| | 5.2 T | reatments Administered | 32 |
|---|---|---|---|
| | 5.2.1 | Investigational Product | 32 |
| | 5.2.2 | Active Comparator | 32 |
| | 5.2.3 | Background Metformin Therapy | 33 |
| | 5.2.4 | Diuretics and Medications for Treatment of Dyslipidemia and | |
| | | Hypertension | |
| | 5.3 S | election and Timing of Dose for Each Patient | |
| | 5.3.1 | 8 | |
| | 5.3.2 | - r | |
| | | Method of Assigning Treatment Groups and Study Drugs | |
| | | linding | |
| | 5.6 C | Concomitant Therapy | 36 |
| | | estrictions | |
| | 5.7.1 | Prior Therapy | 36 |
| | 5.7.2 | | |
| | 5.7.3 | Subject Activity Restrictions | 37 |
| | 5.8 T | reatment Compliance | 37 |
| | 5.9 P | ackaging and Labeling | 37 |
| | 5.9.1 | Run-in Kits | 37 |
| | 5.9.2 | $\varepsilon$ | |
| | 5.9.3 | Glimepiride Kit | 38 |
| | 5.10 S | torage and Accountability | 38 |
| | 5.11 In | rvestigational Product Retention at Study Site | 38 |
| 6 | STUDY | PROCEDURES | 39 |
| | 6.1 In | nformed Consent | 39 |
| | 6.2 S | creening for I/E Criteria | 39 |
| | 6.3 N | Medical History | 39 |
| | 6.3.1 | General Demographics and Characteristics | 39 |
| | 6.3.2 | Diabetes History | 39 |
| | 6.3.3 | Cardiovascular Disease History | 40 |
| | 6.3.4 | Medication History | 40 |
| | 6.4 D | Diet and Exercise Counseling | 40 |
| | 6.5 P | hysical Examination | 40 |
| | 6.6 A | bbreviated Physical Examination | 40 |
| | 6.7 V | 'ital Signs | 41 |
| | 6.8 E | lectrocardiography | 41 |
| | 6.9 C | linical Laboratory Tests | 42 |
| | 6.9.1 | Laboratory Parameters | 42 |

| | 6.9 | 9.2 | Sample Collection, Storage, and Shipping | 42 |
|---|---|---|---|---|
| | | 6.9.2 | | |
| | | <b>.</b> | Control Assessments | |
| | | 6.9.2<br>6.9.2 | J . | |
| | 6.10 | | $\mathcal{E}$ | |
| | | - | and Glucometer Dispensation and Review | |
| | 6.11 | | ensing Run-in Drug | |
| | 6.12 | | and Glucometer Record Review | |
| | 6.13 | _ | ensing Investigational Product | |
| | | 13.1 | Dispensing Bexagliflozin | |
| | | 13.2 | Dispensing Glimepiride | |
| | 6.14 | | Prese Events Assessments | |
| | | 14.1 | Definition of Adverse Events. | |
| | | 14.2 | Eliciting and Reporting AEs | |
| | | 14.3 | Immediately Reportable AEs | |
| | | 14.4 | Pregnancy | |
| | | 14.5 | Procedure for Breaking the Blind | |
| | | 14.6 | Follow-up of Non-Serious AEs | |
| | | 14.7 | Follow-up of Post-Study SAEs | |
| | | 14.8 | Urinary Tract Infections (UTIs) | |
| | | 14.9 | Genital Mycotic Infections (GMIs) | |
| | | 14.10 | Hepatotoxicity | |
| | | 14.11 | Hypoglycemia | |
| | | 14.12 | Diabetic Ketoacidosis (DKA) | |
| | | 14.13 | Major Adverse Cardiovascular Event (MACE) | |
| | | 14.14 | Amputation | |
| | 6.15 | | omitant Medication Assessments | |
| | | | hy-related Quality of Life Assessment | 55 |
| | 6.17 | | oval of Subjects from the Trial or Discontinuation of Investigational | 5.6 |
| | <i>(</i> 10 | | act Administration | |
| 7 | 6.18 | | opriateness of Measurements | |
| 7 | | | | |
| | 7.1 | | ening Period | 5 / |
| | / | 1.1 | Visit V1 (3 days to 3 weeks for metformin-only group and up to 9 weeks for metformin-and-OHA group before run-in period) | 57 |
| | 7.2 | Wast | n-out and Run-in Period (Up to 8 weeks prior to randomization) | |
| | | vv asi<br>2.1 | Wash-out Period (Visits V2 and V3) | |
| | 1.4 | 7.2.1 | · ' | |
| | | 7.2.1 | · • | |

| | 7.2.2 | Run-in Period | 58 |
|---|---|---|---|
| | | 2.2.1 Visit V4 (2 weeks prior to randomization) | |
| | | 2.2.2 Visit V5 (3 to 5 days prior to randomization) | |
| | 7.3 Ti | reatment Period (Day 1 to Week 96) | |
| | 7.3.1 | Visit V6 (Day 1 of Week 1) | 59 |
| | 7.3.2 | Visit V7 (Week 2) | 59 |
| | 7.3.3 | Visit V8 (Week 4) | 59 |
| | 7.3.4 | Visit V9 (Week 6) | 59 |
| | 7.3.5 | Visit V10 (Week 12) | 60 |
| | 7.3.6 | Visit V11 (Week 24) | 60 |
| | 7.3.7 | Visit V12 (Week 36) | 60 |
| | 7.3.8 | Visit V13 (Week 48) | 61 |
| | 7.3.9 | Visit V14 (week 60) | 61 |
| | 7.3.10 | Visit V15 (week 72) | 61 |
| | 7.3.1 | Visit V16 (week 84, off-site phone visit) | 61 |
| | 7.3.12 | 2 Visit V17 (end of treatment, week 96) | 62 |
| | 7.4 V | isit V18 (Exit Visit or Early Termination Visit) | 62 |
| | 7.4.1 | Visit V18 (week 98 or two weeks after the last dose of investigational | |
| | | product is administered or if a subject withdraws consent) | |
| | | iscontinuation of Investigational Product Administration | |
| | | arly Termination Procedures | |
| 8 | - | ΓY CONTROL AND ASSURANCE | |
| 9 | | ED STATISTICAL METHODS | |
| | 9.1 G | eneral Considerations | 65 |
| | 9.2 D | etermination of Sample Size | 65 |
| | 9.3 A | nalysis Populations | 66 |
| | 9.3.1 | Intention-to-Treat Analysis set | 66 |
| | 9.3.2 | Safety Analysis Set | 66 |
| | 9.3.3 | Per Protocol Analysis Set | 66 |
| | 9.4 D | emographics and Baseline Characteristics | 66 |
| | 9.4.1 | Concomitant Medications | 67 |
| | 9.5 Pr | rimary Efficacy Analyses | 67 |
| | 9.5.1 | Hypotheses for the Primary Endpoint | 67 |
| | 9.5.2 | Statistical Methods for Primary Analyses | 67 |
| | 9.5.3 | Analysis of Dropouts Pattern | 68 |
| | 9.6 Se | econdary Efficacy Analyses | 68 |
| | 9.7 O | ther Efficacy Analyses | 69 |
| | 9.8 A | nalysis of Safety | 69 |

| | 9.8 | 8.1 Adverse Events | 69 |
|---|---|---|---|
| | 9.8 | 8.2 Adverse Events of Special Interest | |
| | 9.8 | 8.3 Clinical and Laboratory Events and Analyses | |
| | 9.8 | 8.4 Physical Examination | |
| | 9.9 | Health Related Quality of Life Assessment | |
| | 9.10 | Interim Analysis | |
| | 9.11 | Final Analysis | |
| 10 | ADM | MINISTRATIVE CONSIDERATIONS | 71 |
| | 10.1 | Investigators and Study Administrative Structure | |
| | 10.2 | Institutional Review Board (IRB) or Independent Ethics Committee (IEC Approval | C) |
| | 10.3 | Ethical Conduct of the Study | 71 |
| | 10.4 | Subject Information and Consent | 72 |
| | 10.5 | Subject Confidentiality | |
| | 10.6 | Study Monitoring | 72 |
| | 10.7 | Case Report Forms and Study Records | 73 |
| | 10.8 | Data Monitoring Committee | 73 |
| | 10.9 | Protocol Violations/Deviations | 73 |
| | 10.10 | Access to Source Documentation | 74 |
| | 10.11 | Retention of Data | 74 |
| | 10.12 | Publication and Disclosure Policy | 74 |
| 11 | REFI | ERENCE LIST | 75 |
| LI | ST OI | F IN-TEXT TABLES | |
| | Table | 1. Treatment Groups and Assigned Treatment | 24 |
| | Table | 2. Study Drug Dispensation Schedule | 35 |
| | Table | 3. List of Laboratory Tests | 44 |
| LI: | ST OI | F IN-TEXT FIGURES | |
| | Figure | e 1. Study Design | 20 |
| | Figure | e 2. HbA1c Requirements Prior to Randomization | 23 |
| | Figure | e 3. Glimepiride Dose Up-titration Flow Chart | 26 |
| LI: | ST OI | F APPENDICES | |
| | Appen | ndix 1 Schedule of Events | 7 <i>6</i> |
| | Appen | | |
| | Appen | ndix 3 Sponsor Signatures | 78 |
| | Appen | ndix 4 Investigator's Signature | 79 |

## **SYNOPSIS**

### **Sponsor:**

Theracos Sub, LLC

Name of Finished Product: Bexagliflozin Tablets

Name of Active Ingredient: Bexagliflozin

### **Study Title:**

A Phase 3, Randomized, Double-Blind, Active-Controlled Study to Evaluate the Effects of Bexagliflozin versus Glimepiride in Subjects with Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control by Metformin

Study Number: THR-1442-C-480

Study Phase: 3 Primary Objective:

The primary efficacy objective is to demonstrate that bexagliflozin is non-inferior to glimepiride by evaluating the treatment effect on hemoglobin A1c (HbA1c) reduction at week 60 in subjects whose type 2 diabetes mellitus (T2DM) is inadequately controlled by metformin.

## **Secondary Objectives:**

The key secondary objectives are:

- To evaluate the treatment effect of bexagliflozin vs. glimepiride on the change in body weight in subjects with baseline body mass index (BMI)  $\geq 25 \text{ kg/m}^2$  at week 60
- To evaluate the treatment effect of bexagliflozin vs. glimepiride on the change in systolic blood pressure (SBP) in subjects with baseline SBP  $\geq$  140 mmHg at week 60
- To evaluate the treatment effect of bexagliflozin vs. glimepiride on the difference in proportion of subjects with ≥ 1 severe or documented symptomatic hypoglycemia events over 96 weeks
- To evaluate if bexagliflozin is superior to glimepiride on HbA1c reduction at week 60

#### **Exploratory Objectives:**

- To assess the treatment effect of bexagliflozin vs. glimepiride on the change in the proportion of subjects achieving HbA1c < 7.0% over time
- To assess the treatment effect of bexagliflozin vs. glimepiride on the change in HbA1c over time
- To evaluate the treatment effect of bexagliflozin vs. glimepiride on the change in fasting plasma glucose (FPG) over time
- To assess the treatment effect of bexagliflozin vs. glimepiride on the change in SBP over time
- To assess the treatment effect of bexagliflozin vs. glimepiride on the change in body weight over time
- To assess the treatment effect of bexagliflozin vs. glimepiride on the difference in proportion of subjects with ≥ 1 severe or documented symptomatic hypoglycemia events over time

 Version 3.0 (Global)

### **Safety Objectives:**

- To compare the effects of bexagliflozin vs. glimepiride on the incidence of adverse events of interest. Adverse events of interest are urinary tract infections including urosepsis and pyelonephritis, genital mycotic infections, diuretic effects including hypovolemia, hypotension episodes, hypoglycemia, hepatotoxicity, major adverse cardiovascular events (MACE), falls and fractures, malignancies, hypersensitivity reactions, acid-base disorders including diabetic ketoacidosis, and renal failure events.
- To compare the effects of bexagliflozin vs. glimepiride on general safety assessments including treatment emergent adverse events, clinical laboratory events, 12-lead electrocardiograms (ECG) parameters, physical examinations, vital signs including orthostatic blood pressure, and use of concomitant medications

# **Other Objectives:**

• To compare the effects of bexagliflozin vs glimepiride on health-related quality of life using a validated instrument EQ-5D-3L.

## **Study Design:**

THR-1442-C-480 is a phase 3, multi-center, randomized, double-blind, parallel-group study to evaluate the efficacy and safety of bexagliflozin versus glimepiride in subjects T2DM is inadequately controlled by metformin. A total of420 subjects are planned to be randomized in a ratio of 1:1 to receive once daily treatment of active bexagliflozin with placebo glimepiride (Group 1) or placebo bexagliflozin with active glimepiride (Group 2) for 96 weeks in an outpatient setting. Active treatment in Group 1 will be bexagliflozin tablets, 20 mg. Active treatment in Group 2 will be glimepiride capsules, 2, 4, or 6 mg. At the time of screening, subjects will be taking metformin only (metformin-only) or metformin in addition to no more than one additional oral hypoglycemic agent (metformin-and-OHA). Study subjects will continue receiving open-labeled metformin background medication during the entire study.

The main eligibility criteria include 1) male or female subjects with T2DM and 2) screening HbA1c between 7.0% and 10.5% (inclusive) for subjects who are metformin-only treated, or screening HbA1c between 6.5% and 10.0% (inclusive) for subjects who are metformin-and-OHA treated.

All eligible subjects must have taken metformin at a stable dose of  $\geq 1500$  mg/day for at least 8 weeks prior to screening. Subjects who are metformin-and-OHA treated must be willing to undergo a 6-week wash-out of the non-metformin OHA prior to the start of a 2 week run-in period. During the wash-out, subjects will discontinue non-metformin OHA and continue taking metformin at the dose and frequency taken at screening.

All eligible subjects who are metformin-only treated or have completed the 6-week wash-out period will start a 2-week single-blind run-in period. During the run-in, subjects will receive placebo bexagliflozin and placebo glimepiride. Subjects who meet all inclusion criteria and no exclusion criteria prior to randomization will be eligible for randomization and receive


investigational products.

During the treatment period, glimepiride will be provided in three dose levels: 2 mg, 4 mg, and 6 mg. Placebo glimepiride will also be provided in three dose levels: placebo for 2 mg, placebo for 4 mg, and placebo for 6 mg. Subjects will receive the starting dose of glimepiride, 2 mg or placebo. Subjects who meet protocol-specified glycemic criteria will undergo up-titration of the glimepiride dose at weeks 2, 4, and 6. The dose will be increased to the next dosing level if during the proceeding 2 weeks:  $(1) \ge 50\%$  of fasting SMBG measurements > 110 mg/dL and (2) no severe or documented symptomatic hypoglycemia events. Subjects assigned to receive placebo glimepiride, will receive mock titrations of glimepiride at weeks 2, 4, and 6 based on the same glycemic criteria. No dose changes of glimepiride will occur after 6 weeks of treatment.

Each subject will be instructed to return to the clinic at weeks 0, 2, 4, 6, 12, 24, 36, 48, 60, 72, 84 (off-site phone visit) and 96 for efficacy assessment and safety monitoring. Subjects will return to the clinic for a follow-up exit visit at week 98 or 2 weeks after last dose of study drug if subjects early terminate prior to week 96.

During the study, a Data and Safety Monitoring Board (DSMB) will review the unblinded data periodically and may recommend an early termination of the trial for safety reasons. In the event of administrative changes or other related reasons, the sponsor reserves the rights to terminate the study early. There will be no interim analysis; final statistical analysis will be performed after all subjects complete the study.

#### Study Population and Main Eligibility Criteria:

A total of 420 eligible subjects are planned for this study. The study population will comprise:

- 1. Male or female adult subjects  $\geq$  18 years of age
- 2. If subjects are female of childbearing potential, subjects must be negative on the urine pregnancy test and agree to abstain from coitus or use contraception during the entire study to avoid any possible pregnancy
- 3. Subjects who are in one of the two categories:
  - a. Metformin-only treated: receive ≥ 1500 mg/day metformin only for at least 8 weeks prior to screening or
  - b. Metformin-and-OHA treated: receive ≥ 1500 mg/day metformin for at least 8 weeks prior to screening and ≥ 14 days of 1 additional oral hypoglycemia agent (OHA) in the 8 weeks prior to screening.
- 4. Subjects with a diagnosis of T2DM with HbA1c levels between 7.0% and 10.5% (inclusive) at screening if metformin-only treated or with HbA1c levels between 6.5% and 10.0% (inclusive) at screening if metformin- and-OHA treated
- 5. Subjects with a body mass index (BMI)  $\leq$  45 kg/m<sup>2</sup> at screening
- 6. If applicable, taking stable doses of treatment for dyslipidemia and/or hypertension for 30 days prior to screening. Subjects do not need to be treated for dyslipidemia or hypertension to be eligible for the study


7. Subjects who are willing and able to return for all clinic visits and to complete all study-required procedures, including self-monitoring blood glucose (SMBG) measurements

Prior to randomization, all subjects must:

- 8. Maintain adequate glycemic control during the washout and run-in periods (fasting plasma glucose values are not  $\geq 250 \text{ mg/dL}$  on consecutive days)
- 9. Have an HbA1c between 7.0% and 10.5% (inclusive) at Visit V5
- 10. Adhere to the investigational product administration requirements as evidenced by missing no more than 2 placebo run-in medication doses of any kind

#### Test Products, Dose, and Mode of Administration:

Once daily oral administration of bexagliflozin and glimepiride

- Group 1: bexagliflozin tablets, 20 mg, and glimepiride capsules, placebo
- Group 2: bexagliflozin tablets, placebo, and glimepiride capsules, 2 mg, 4 mg or 6 mg

#### **Duration of Treatment:**

Eligible subjects will receive a total treatment duration of 98 weeks including 2 weeks of run-in medications and 96 weeks of investigational products.

### **Efficacy Assessments:**

## Primary efficacy assessment:

• Change in HbA1c from baseline at week 60

## Secondary efficacy assessments:

- Change in body weight in subjects with baseline body mass index (BMI)  $\geq$  25 kg/m<sup>2</sup> at week 60
- Change in SBP in subjects with baseline SBP  $\geq$  140 mmHg from baseline at week 60
- Difference in proportion of subjects with ≥ 1 severe or documented symptomatic hypoglycemia events over 96 weeks
- Change in HbA1c from baseline at week 60

## Other efficacy endpoints:

- Change in proportion of subjects achieving HbA1c < 7.0% over time
- Change in body weight over time
- Change in FPG over time
- Change in SBP over time
- Change in HbA1c over time
- Difference in proportion of subjects with ≥ 1 severe or documented symptomatic hypoglycemia events over time


#### Safety Endpoints:

Adverse events, including adverse events of special interest (genital and urinary tract
infections, diuretic effects, hepatotoxicity, MACE, hypoglycemia, fractures, malignancy,
hypersensitivity reactions, hypotensive episodes, acid-base disorders, and renal failure
events)

- Laboratory testing, including hematology, serum chemistry, and urinalysis
- Physical examination
- 12-lead ECG
- Vital signs
- Concomitant medication use

#### Other Assessment:

Health-related quality of life instrument EQ-5D-3L

#### **Statistical Methods:**

The primary hypothesis is that bexagliflozin is non-inferior to glimepiride by evaluating the treatment effect on HbA1c reduction at week 60 in combination with metformin. The noninferiority margin for mean change from baseline at week 60 in HbA1c comparing bexagliflozin group with glimepiride group will be 0.35%. Superiority will be declared without additional statistical testing when the upper bound of the 95% CI for difference in change from baseline at week 60 in HbA1c comparing bexagliflozin group with glimepiride group is less than 0. The treatment difference will be examined by using a mixed model repeated measures (MMRM) analysis of covariance model (ANCOVA). The model will include treatment, visit, treatment-by-visit interaction and randomization stratification factors as the fixed effects terms and the baseline HbA1c value as a fixed effect covariate. Least squares mean treatment differences between the bexagliflozin group and the comparator group at week 60 in change from baseline will be estimated from the model. An unstructured covariance will be used to model the within-subject correlation. If the model with the unstructured covariance structure does not converge, an autoregressive(1) covariance structure will be used. HbA1c values obtained after the start of rescue medication will not be excluded from this primary analysis. Primary endpoint will be analyzed on both intention-totreat (ITT) and per protocol (PP) analysis sets.

The MMRM model is one approach to obtain treatment effect estimates in the presence of missing data. As sensitivity analyses for missing data, the following will be performed on both ITT and PP analysis sets:

- 1. Missing data will be imputed via multiple imputations, following which the MMRM will be repeated on the complete datasets with results combined across complete datasets using standard multiple imputation techniques; HbA1c values collected after the start of rescue medication will not be excluded.
- 2. Missing data will be imputed via LOCF, following which the MMRM will be repeated; HbA1c values collected after the start of rescue medication will be considered missing.
- 3. HbA1c values collected after the start of rescue medication will be considered missing,


and the MMRM analyses will be re-performed.

The effects of bexagliflozin on the changes from baseline at week 60 in body weight and systolic blood pressure, the difference in the proportion of subjects with  $\geq 1$  severe or documented symptomatic hypoglycemia events over 96 weeks and the change in HbA1c from baseline at week 60 will be tested as key secondary endpoints and will be analyzed in a hierarchical testing strategy and only if the primary objective is met. Similar to the primary endpoint, ANCOVA models will be used for the continuous secondary endpoints and logistic regression model will be used for the binary endpoint. A hierarchical testing strategy will be followed to preserve experiment-wide alpha at 0.05:

- 1. Superiority test of the change in body weight in subjects with baseline BMI  $\geq$  25 kg/m<sup>2</sup> in the bexagliflozin group vs. the glimepiride group at week 60
- 2. Superiority test of the change in systolic blood pressure (SBP) in subjects with baseline SBP ≥ 140 mmHg in the bexagliflozin group vs. the glimepiride group at week 60
- 3. Superiority test of the difference in proportion of subjects with ≥ 1 severe or documented symptomatic hypoglycemia event in the bexagliflozin group vs. the glimepiride group over 96 weeks

Additional effects of bexagliflozin versus glimepiride on the changes in HbA1c, FPG, SBP, body weight, the proportion of subjects who reach an HbA1c < 7%, and the proportion of subjects with  $\ge 1$  severe or documented symptomatic hypoglycemia events over time, as well as the general safety in subjects with T2DM, will be analyzed as exploratory efficacy endpoints. These endpoints are considered exploratory and will not be adjusted for multiplicity.

For the primary efficacy endpoint, a minimum of 172 subjects are needed in each treatment arm to detect non-inferiority of bexagliflozin to glimepiride with respect to the change in HbA1c from baseline at week 60 by a margin of 0.35%, assuming an estimated pooled standard deviation of 1.0%. This estimation is based on a one-sided t-test with 90% power at a 0.025 level of significance. To allow for an estimated 18.0% dropout rate, 210 patients will be randomized in each treatment arm, and the total sample size will be 420 subjects for this study.

Statistical analyses and summaries will be performed using  $SAS^{\circledR}$  software (SAS Institute, Cary, NC).


## LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

ADA American Diabetes Association

AE adverse event

ALB albumin

ALT alanine aminotransferase
ANCOVA analysis of covariance
AST aspartate aminotransferase

ATC Anatomic Therapeutic Chemical classification

BMI body mass index
BP blood pressure
BUN blood urea nitrogen

CEC cardiovascular endpoint committee

CFR Code of Federal Regulations

CI confidence interval CRF case report form

CRO contract research organization

DKA diabetic ketoacidosis
CYP cytochrome P450
DPP4 dipeptidyl peptidase-4

DSMB data and safety monitoring board

ECG electrocardiogram

eGFR estimating glomerular filtration rate

FPG fasting plasma glucose GCP Good Clinical Practice

GI gastrointestinal

GLP-1 glucagon-like peptide-1 GMI genital mycotic infection

h hour

HbA1c hemoglobin A1c

HBsAg hepatitis B surface antigen

Hct hematocrit HCV hepatitis C virus

HDL-C high density lipoprotein cholesterol

HDPE high-density polyethylene

Hgb hemoglobin

HIV human immunodeficiency virus

ICH International Conference on Harmonisation

Bexagliflozin Tablets Clinical Trial Protocol: THR-1442-C-480

IEC independent ethics committee

IND Investigational New Drug application IRAE immediately reportable adverse event

IRB institutional review board

ITT intention-to-treat

IWRS Interactive Web Response System
LDL-C low density lipoprotein cholesterol
LOCF last observation carried forward
MACE major adverse cardiovascular event
MCH mean corpuscular hemoglobin

MCHC mean corpuscular hemoglobin concentration

MCV mean corpuscular volume

MDRD modification of diet in renal disease

MedDRA medical dictionary for regulatory activities

MI myocardial infarction

MMRM mixed model repeated measures
MODY maturity—onset diabetes of the young

N number of subjects

NYHA New York Heart Association
OHA oral hypoglycemic agent

PO per oral PP per protocol

PR time from the beginning of the P wave to the beginning of the QRS

complex in electrocardiogram

ORS QRS complex is a name for the combination of three of the graphical

deflections seen on a typical electrocardiogram

corrected QT interval is a measure of the time between the start of the Q

wave and the end of the T wave in the heart's electrical cycle

RBC red blood cell (count)
SAE serious adverse event
SBP systolic blood pressure
SD standard deviation

SGLT2 sodium glucose cotransporter 2 SMBG self-monitored blood glucose SOP standard operating procedure

SU sulfonylurea

SUSAR serious and unexpected suspected adverse event

T2DM type 2 diabetes mellitus

Bexagliflozin Tablets Clinical Trial Protocol: THR-1442-C-480

TC total cholesterol

TEAE treatment emergent adverse event

TG triglycerides

TZD thiazolidinedione

UACR urine albumin to creatinine ratio
UADR unexpected adverse drug reaction

UGE urinary glucose excretion
ULN upper limit of normal
UPT urinary pregnancy test
UTI urinary tract infections
WBC white blood cell (count)

WHO-DD World Health Organization Drug Dictionary

WOCBP women of childbearing potential

## 1 INTRODUCTION

Type 2 diabetes mellitus (T2DM) is one of the leading causes of morbidity and mortality worldwide, affecting an estimated 415 million people in 2015. Approximately 187 million of those affected are thought to be unaware of their condition and over 80% reside in low- and middle-income countries (IDF 2015).

# 1.1 Type 2 Diabetes Mellitus

T2DM is the predominant form of diabetes and accounts for at least 90% of all diabetes cases, which is characterized by insulin resistance and relative or absolute insulin insufficiency. Despite the availability of several classes of therapeutics, the number of people with diabetes is projected to increase by nearly 55% to over 642 million adults by 2040 (IDF 2015). Among the debilitating consequences of T2DM are peripheral neuropathy, retinopathy, renal failure, peripheral ischemia and exacerbations of cardiovascular disease, which result in blindness, amputation, dialysis and death.

T2DM is a disease strongly linked to increased body fat mass in the majority of cases (Schwartz, Fabricatore et al. 2012). Weight loss has been shown to improve glycemic control and to reduce the severity of diabetes-associated comorbidities, supporting the view that antidiabetic agents that promote weight loss may be particularly beneficial for the treatment of the disease (Look, Wing et al. 2013; Scheen and Van Gaal 2014). Several classes of agents are available for treating T2DM, including insulin and its secretagogues such as, sulfonvlureas (SU), PPARy agonists, biguanides, alpha glucosidase inhibitors, glucagon-like peptide 1 (GLP-1) receptor agonists, sulfonylureas, meglitinides, dipeptidyl peptidase 4 (DPP4) inhibitors, and sodium glucose linked transporter 2 inhibitors (SGLT2i). Metformin is the first line medication for treating T2DM; however, as T2DM progresses over time, metformin monotherapy is not able to adequately manage hyperglycemia. T2DM patients often receive more than one antidiabetic medication after an initial treatment period of metformin monotherapy. SU are considered second-line therapy for T2DM in clinical practice and are often prescribed with metformin as a combination therapy for treating T2DM. SU can reduce the risk of long-term microvascular complications via effective glycemic control; however, common side effects include weight gain and increased risk of hypoglycemia. The durability of SU treatment can be reduced due to loss of β-cell function as T2DM progresses over time.

The rapid growth rate in the incidence of T2DM has led to an increasing recognition that additional therapeutics are needed to provide safe and effective reductions of elevated plasma glucose levels. New agents to treat T2DM, either as monotherapy or add-on therapy to other anti-diabetic medications, would ideally treat hyperglycemia and avoid common side effects of currently available agents, such as weight gain, gastrointestinal disturbance, and hypoglycemia.

The renal Na+/glucose transport protein SGLT2 actively transports extracellular glucose into cells using the driving energy of the transmembrane electrochemical potential for sodium ions. Individuals with disruptions in *SLC5A2*, the gene encoding SGLT2, exhibit prominent


glucosuria in the absence of significant co-morbidities (van den Heuvel, Assink et al. 2002; Santer, Kinner et al. 2003). The excretion of glucose in the urine of diabetic subjects in amounts comparable to or greater than that seen in individuals harboring loss of functions mutations in *SLC5A2* has the potential to improve fasting and postprandial hyperglycemia without increasing insulin secretion, causing weight gain, or inducing hypoglycemia. Several SGLT2 inhibitors have demonstrated these clinical benefits, as well as sustained weight loss when used as a mono-therapy or in combination with other oral anti-diabetic medications including insulin (Nauck 2014; Seufert 2015).

# 1.2 Bexagliflozin for the Treatment of Type 2 Diabetes Mellitus

Bexagliflozin is a candidate oral hypoglycemic agent (OHA) that is a potent and highly specific inhibitor of SGLT2. It was identified following a synthetic program aimed at creating molecules with high selectivity and potency for SGLT2 (Zhang, Welihinda et al. 2011). Bexagliflozin has been shown to cause dose-dependent increases in urinary glucose excretion (UGE) in humans, rats, dogs and monkeys and to reduce HbA1c in animal models of T2DM as well as in diabetic subjects. The safety and efficacy of bexagliflozin capsules, 20 mg, were evaluated in a 96-week study that measured reduction in hemoglobin A1c as the primary endpoint. Adverse event incidences, particularly for urinary tract infection (UTI) and genital mycotic infection (GMI), were similar between placebo and active agent cohorts. Details of the pharmacology, efficacy, and safety assessments are described in the Investigator's Brochure.

### 2 STUDY OBJECTIVES

# 2.1 Primary Objective

The primary efficacy objective of this trial is to demonstrate that bexagliflozin is non-inferior to glimepiride by evaluating the treatment effect on HbA1c reduction at week 60 in subjects whose T2DM is inadequately controlled by metformin.

# 2.2 Key Secondary Objectives

- To evaluate the treatment effect of bexagliflozin vs. glimepiride on the change in body weight in subjects with baseline body mass index (BMI)  $\geq 25 \text{ kg/m}^2$  at week 60
- To evaluate the treatment effect of bexagliflozin vs. glimepiride on the change in systolic blood pressure (SBP) in subjects with baseline SBP ≥ 140 mmHg at week 60
- To evaluate the treatment effect of bexagliflozin vs. glimepiride on the difference in proportion of subjects with ≥1 severe or documented symptomatic hypoglycemia events over 96 weeks
- To evaluate if bexagliflozin is superior to glimepiride on HbA1c reduction at week 60

# 2.3 Exploratory Objectives

- To assess the treatment effect of bexagliflozin vs. glimepiride on the change in the proportion of subjects achieving HbA1c < 7.0% over time
- To assess the treatment effect of bexagliflozin vs. glimepiride on the change in HbA1c over time
- To assess the treatment effect of bexagliflozin vs. glimepiride on the change in fasting plasma glucose (FPG) over time
- To assess the treatment effect of bexagliflozin vs. glimepiride on the change in SBP over time
- To assess the treatment effect of bexagliflozin vs. glimepiride on the change in body weight over time
- To assess the treatment effect of bexagliflozin vs. glimepiride on the difference in proportion of subjects with ≥ 1 severe or documented symptomatic hypoglycemia events over time

#### **Safety Objectives:**

- To compare the effects of bexagliflozin vs. glimepiride on the incidence of adverse events of interest. Adverse events of interest are urinary tract infections including urosepsis and pyelonephritis, genital mycotic infections, diuretic effects including hypovolemia, hypotension episodes, hypoglycemia, hepatotoxicity, major adverse cardiovascular events (MACE), falls and fractures, malignancies, hypersensitivity reactions, acid-base disorders including diabetic ketoacidosis, and renal failure events.
- To compare the effects of bexagliflozin vs. glimepiride on general safety assessments including treatment emergent adverse events, clinical laboratory events, 12-lead


electrocardiograms (ECG) parameters, physical examinations, vital signs including orthostatic blood pressure, and use of concomitant medications

# **Other Objectives:**

• To compare the effects of bexagliflozin and glimepiride on health-related quality of life using a validated instrument EQ-5D-3L

#### 3 INVESTIGATIONAL PLAN

## 3.1 Overall Study Design and Plan

THR-1442-C-480 is a phase 3, multi-center, randomized, double-blind, parallel-group study and aims to demonstrate that bexagliflozin is non-inferior to glimepiride as add-on therapy in subjects whose T2DM is not adequately controlled by metformin treatment. The primary efficacy endpoint is the change in HbA1c from baseline at week 60. The study will enroll T2DM patients who are treated with only metformin (metformin-only) or who are treated with metformin and one additional oral hypoglycemic agent (metformin-and-OHA)

All subjects must have taken metformin at a stable dose of  $\geq$  1500 mg/day for  $\geq$  8 weeks prior to screening. Subjects can be eligible for the metformin-only treated group if they have received < 14 days of any other antidiabetic medications in the 8 weeks prior to screening. Subjects can be eligible for the metformin-and-OHA treated group if they have received  $\geq$  14 days of no more than 1 other OHA in the 8 weeks prior to screening; subjects taking any other antidiabetic medication (in addition to metformin and the 1 OHA) for < 14 days in the 8 weeks prior to screening are allowed.

A total of 420 subjects who meet all the inclusion criteria, none of the exclusion criteria, and who consent to participate in the study, are eligible for study enrollment. Metformin-and-OHA treated subjects will undergo a 6-week washout of the non-metformin OHA prior to the start of run-in. Subjects who complete the 2-week run-in and who meet all eligibility criteria will be randomized in a 1:1 ratio to receive once daily double-blind treatment of either active bexagliflozin tablets with placebo glimepiride capsules (Group 1) or placebo bexagliflozin tablets and active glimepiride capsules (Group 2). Active treatment in Group 1 will be bexagliflozin tablets, 20 mg. Active treatment in Group 2 will be glimepiride capsules, 2, 4 or 6 mg. Study subjects will continue receiving open-labeled metformin background medication during the entire study at a stable dose and frequency. The treatment period will last 96 weeks and be conducted in an outpatient setting (Figure 1).



Figure 1. Study Design

# 3.2 Rationale for Study Design and Control Group

# 3.2.1 Rationale for Background Medication and Active Comparator

Metformin is the most commonly prescribed OHA and is recommended as first-line therapy for the treatment of T2DM. However, subjects who have T2DM often require multiple anti-


diabetic medications for glycemic control. Sulfonylureas are often prescribed with metformin as a combination therapy for treating T2DM. Sulfonylureas can reduce the risk of long-term microvascular complications via effective glycemic control. Yet, common side effects of sulfonylureas include weight gain and increased risk of hypoglycemia. Glimepiride is one of the most commonly prescribed second-generation sulfonylureas. Thus, it is an appropriate active comparator in the subject population studied during the treatment period (96 weeks).

Bexagliflozin is an SGLT2 inhibitor developed for the treatment of T2DM that reduces hyperglycemia via an insulin-independent pathway of inhibiting glucose re-uptake and promoting urinary glucose excretion. Individuals treated with metformin and with inadequate glycemic control have reduced HbA1c, reduced body weight, and less incidence of hypoglycemia when treated with approved SGLT2 inhibitors canagliflozin, dapagliflozin or empagliflozin. Thus T2DM subjects on metformin therapy with inadequate glycemic control may benefit from combination treatment with bexagliflozin.

## 3.2.2 Rationale for the Study Design

THR-1442-C-480 is designed to assess the non-inferiority of bexagliflozin to glimepiride as add-on therapy to metformin for glycemic control in T2DM subjects.

To assess the effect of bexagliflozin or glimepiride in addition to an effective dose of metformin background therapy, all subjects must be taking a stable dose of  $\geq 1500$  mg metformin daily for at least 8 weeks prior to screening. If a potential subject has taken < 1500 mg/day metformin, alone or in combination with 1 other OHA, the subject can enter screening once the dose of metformin has been be increased to at least 1500 mg/day for at least 8 weeks. Changes in the dose of metformin will not be permitted at any time during the study.

To exclude the possibility that OHAs other than metformin taken prior to study enrollment might influence study outcomes, subjects who are metformin-and-OHA treated will undergo a 6-week wash-out of the non-metformin OHA prior to the start of run-in. During the wash-out, subjects will discontinue non-metformin OHA and continue taking metformin at the dose and frequency taken at screening.

Diet and exercise counseling will be provided to all participating subjects to reduce risks of worsening diabetic conditions. A monitoring plan and criteria to initiate rescue medications are included in the protocol to prevent prolonged hyperglycemia.

Reduction in HbA1c directly reflects improvement in glycemic control and is considered a well-validated surrogate for the long-term microvascular complications of diabetes mellitus. Therefore the primary endpoint of change in HbA1c measurement from baseline at 60 weeks will reflect the long-term effects of bexagliflozin compared with glimepiride.

#### 3.2.3 Rationale for the Dose Selection

Bexagliflozin produces a dose-dependent, saturable increase in UGE in healthy volunteers and diabetic subjects. Population pharmacodynamic modeling has indicated that


bexagliflozin doses of 20 mg result in 90% of the maximal UGE. In a long term treatment study, daily administration of 20 mg bexagliflozin was found to reduce HbA1c by 0.79% compared to placebo at week 24. The treatment benefit was observed to improve to 1.02% at week 96. FPG reduction, weight loss, and decreased systolic and diastolic blood pressures were also observed following 96 weeks of treatment. In addition, adverse events (AEs), particularly those involving UTI and GMI, were found to be similar between placebo and active agent cohorts. To evaluate the safety and efficacy of bexagliflozin for the treatment of subjects with T2DM, bexagliflozin tablets, 20 mg will be administered in this trial. Sulfonylureas are known to increase the risk of hypoglycemia. To control hyperglycemia and minimize hypoglycemia, subjects randomized to Group 2 will start with glimepiride at 2 mg daily and undergo dose up-titration based on protocol-specific criteria during the first 6 weeks of the study (Section 3.3.2.1).

#### 3.3 Research Methods and Procedures

#### 3.3.1 Wash-out and Run-in Period

Subjects who are metformin-and-OHA treated will undergo a 6-week wash-out of the non-metformin OHA prior to the start of a 2 week run-in period. During the wash-out, subjects will discontinue non-metformin OHA and continue taking metformin at the dose and frequency taken at screening.

At the start of the washout, metformin-and-OHA treated subjects will receive diet and exercise counseling as well as instructions on contacting the clinic in the event of hyperglycemia, hypoglycemia, or symptoms that may suggest ketoacidosis. Study subjects will be provided with a glucometer and instructions for its daily use. Two weeks after the start of the wash-out period, each subject will participate in a phone interview visit with study staff for SMBG data review and general safety evaluation. Subjects who remain eligible at the end of the washout period will begin a two-week run-in period.

Metformin-only treated subjects will not undergo washout; they will proceed directly to the start of run-in. At the start of the run-in period, metformin-only treated subjects will receive diet and exercise counseling as well as instructions on contacting the clinic in the event of hyperglycemia, hypoglycemia, or symptoms that may suggest ketoacidosis. Metformin-and OHA treated subjects will receive this information at the start of the washout period. At the start of run-in, metformin-only treated subjects will be provided with a glucometer and instructions for its daily use.

All eligible subjects who are metformin-only treated or have successfully completed the 6-week wash-out period will start a 2-week single-blind run-in period. During the run-in, subjects will receive placebo bexagliflozin and placebo glimepiride. Bexagliflozin tablets, placebo, will be taken once daily in the morning prior to the first meal and glimepiride capsules, placebo, will be taken once daily in the morning with the first meal; the medications should be taken with water. Metformin dose and frequency will remain unchanged from time of screening throughout the course of the study.

Subjects will <u>not</u> be eligible for randomization if during the run-in period they:


- 1. have fasting blood glucose values  $\geq 250 \text{ mg/dL}$  on two or more consecutive days,
- 2. omit more than 2 placebo run-in medication doses of any kind,
- 3. are deemed inappropriate for the study by the investigator, or
- 4. have an HbA1c value < 7.0% or > 10.5% at visit V5. The glycemic control requirement based on HbA1c values is outlined in Figure 2.



Figure 2. HbA1c Requirements Prior to Randomization

Changes in the dose of treatment for dyslipidemia or hypertension will not be permitted during the screening and run-in periods.

If a change in treatment for hypertension or dyslipidemia is deemed necessary by the investigator for the well-being of the study subject during the screening or washout periods, the subject will be considered as screen failed and discontinue study activities; the subject may be re-screened as a new subject after the clinical condition and treatment regimen have not changed for at least 30 days. When re-screening, a new subject number will be assigned and all screening activities, including informed consent, and assessments will be performed.

If a change in treatment for hypertension or dyslipidemia is deemed necessary by the investigator for the well-being of the study subject during the run-in period, the subject will be considered as screen failed and discontinue study activities; there will be no opportunity to re-screen for subjects who have started run-in or failed screening.

#### 3.3.2 Treatment Period

The double-blind treatment period will start at randomization and last 96 weeks. A total of 420 subjects of 210 subjects per group will be randomized in a 1:1 ratio to the two groups as shown in Table 1.


Table 1. Treatment Groups and Assigned Treatment

| Treatment Group | Treatment |
|---|---|
| 1 | Bexagliflozin tablets, 20 mg, (once daily P.O.)<br>Glimepiride capsules, placebo, (once daily P.O.) |
| 2 | Bexagliflozin tablets, placebo, (once daily P.O.)<br>Glimepiride capsules, 2, 4 or 6 mg, (once daily P.O.) |

Randomization will be stratified by HbA1c at Visit V5 ( $\leq$  8.5% vs. > 8.5%), treatment background (metformin-only vs. metformin-and-OHA), and baseline estimated glomerular filtration rate (eGFR) at screening visit (V1) (eGFR  $\geq$  90 vs. < 90 and  $\geq$  60 mL/min/1.73 m<sup>2</sup>). At the start of the treatment period, each subject will be provided with bexagliflozin tablets, glimepiride capsules, dosing instructions, and a glycemic control diary in which to record SMBG measurements. Symptoms and blood sugars related to the occurrence of hyperglycemia, hypoglycemic events or symptoms that may suggest ketoacidosis will be recorded. Bexagliflozin tablets, 20 mg or placebo, will be orally administered once daily prior to the first meal; glimepiride capsules, 2, 4, or 6 mg or placebo, will be taken once daily with the first meal. Background medication metformin shall be taken at an unchanged dose and frequency taken at screening throughout the entire study.

Each subject will be instructed to return to the clinic at weeks 0, 2, 4, 6, 12, 24, 36, 48, 60, 72, 84 (off-site phone visit) and 96 for efficacy assessment and safety monitoring, including review of adverse events and concomitant medication, vital signs, ECG, physical examination, and blood and urine specimen collections. On the day of a clinic visit at which blood samples are scheduled to be collected, approximately 10 hours (h) fasting must be confirmed prior to blood draw. On the day of the scheduled clinic visits at which there is fasting and blood is to be drawn, administration of bexagliflozin shall be withheld until after blood is drawn and taken with water at the clinic or home prior to the first meal; glimepiride shall be withheld and taken with the first meal of the day.

Subjects will return to the clinic for a follow-up exit visit at week 98 or 2 weeks after the last dose of study drugs if subjects early terminate prior to week 96. Following the exit visit, subjects will be advised to see their primary physician to undergo treatment to control their diabetes.

#### 3.3.2.1 Glimepiride Dose Titration

During the treatment period, glimepiride will be provided in three dose levels: 2 mg, 4 mg, and 6 mg. Glimepiride placebo will also be provided.

#### Weeks 0 to 6

Subjects will receive the starting dose of glimepiride at 2 mg or placebo at week 0 (V6).

At weeks 2, 4 and 6 (scheduled visits V7, V8 and V9, respectively), subjects will return to the clinic for the assessment of glimepiride dose up-titration and safety evaluation. If subjects


meet the following glycemic criteria in the preceding 2 weeks, glimepiride dose will be increased to the next level.

- 1.  $\geq$  50% of documented fasting SMBG measurements  $\geq$  110 mg/dL (6.1mmol/L)
- 2. no severe or documented symptomatic hypoglycemia events

Subjects assigned to receive placebo glimepiride, will receive mock titrations of glimepiride at weeks 2, 4, and 6 based on the same glycemic criteria.

In case of persistent hyperglycemia [more than 3 consecutive daily, fasting SMBG measures ≥ 270 mg/dL (15mmol/L)] during the treatment period, subjects should contact the clinic and schedule the up-titration visit(s) early to receive the next higher dose of glimepiride.

During weeks 0 to 6, each up-titration visit should be conducted no more than 2 weeks after the prior visit. Visits V6 and V9 will always occur at week 0 and week 6, respectively.

In the case that subjects experience persistent hyperglycemia and up-titration visits are scheduled early, if more than two weeks elapse between scheduled visits or an up-titration is needed between scheduled visits, an unscheduled visit with the same study procedures and tests as the previous scheduled visit will be conducted during the unscheduled visit.

If subjects do not meet up-titration glycemic criteria, subjects will continue glimepiride at the same dose prescribed to them at previous visit. The up-titration schema is demonstrated in Figure 3.

#### Weeks 7 to 96

No dose changes in glimepiride will occur after 6 weeks of treatment. Subjects will continue receiving glimepiride at the unchanged dose, time, and frequency prescribed to them at week 6.

Down-titration of glimepiride is not allowed during the entire study.

At the discretion of the investigator, subjects who experience recurring symptomatic hypoglycemia or any severe episode of hypoglycemia during the treatment period can discontinue study drug.




<sup>\*</sup>If subjects have persistent hyperglycemia [more than 3 consecutive daily, fasting SMBG measures  $\geq$  270 mg/dL (15mmol/L)], subjects should contact the clinic and schedule the up-titration visit(s) early to receive the next higher dose of glimepiride

Figure 3. Glimepiride Dose Up-titration Flow Chart

#### 3.3.3 Glycemic Control Monitoring

#### 3.3.3.1 Wash-out Period and Placebo Run-in Period

During the wash-out and placebo run-in period, subjects will be instructed to determine SMBG daily after fasting overnight for a minimum of 10 h. Subjects should contact the clinic if any fasting glucose value is  $\geq 250$  mg/dL (13.9 mmol/L), and the investigator will determine whether the participant should attempt to improve diet and exercise to maintain glycemic control or if the participant must withdraw from the study and initiate a more intense pharmacological regimen for glucose control.

A subject will be excluded from further participation if his fasting blood glucose is  $\geq 250$  mg/dL prior to randomization on 2 or more consecutive days. Subjects with clinical signs or symptoms of severe hyperglycemia during the wash-out or run-in periods, including weight loss, blurred vision, increased thirst, increased urination, or fatigue, should also be excluded.

#### 3.3.3.2 Treatment Period

During the treatment period, subjects will be advised to continue daily, fasting SMBG measurements. Subjects should contact the clinic if any fasting SMBG is  $\geq$  270 mg/dL (15 mmol/L) from week baseline to week 6,  $\geq$  240 mg/dL (13.3 mmol/L) after week 6 to week 12, or  $\geq$  200 mg/dL (11.1 mmol/L) after week 12. Blood glucose values collected via SMBG will be evaluated at study visits by the investigator. In addition, hyperglycemia will be monitored by FPG at scheduled visits.


If hyperglycemia is identified through SMBG or FPG measurements, the investigator will determine whether the subject has fasted for a minimum of 10 h prior to the morning blood draw to ensure that the SMBG or FPG value is truly a fasting sample. If proper fasting has not occurred, the subject will be asked to return for a repeat blood test within a week.

During the treatment period, hyperglycemia should be managed first with diet and exercise counseling. If hyperglycemia continues after diet and exercise counseling, the investigator should intensify medical therapy if it is necessary for the well-being of the subject. Options for intensification of medical therapy will vary during the study, including up-titration of glimepiride dose (weeks 0-6) and addition of rescue medication (see below, *Intensification of Medical Therapy for Hyperglycemia*).

#### 3.3.3.3 Intensification of Medical Therapy for Hyperglycemia

During the entire treatment period, a review of diet and exercise counseling is suggested prior to prescription of rescue medication in the absence of specific medical indications for rescue medication.

Intensification of medical therapy for hyperglycemia is suggested during the treatment period if, after diet and exercise counseling, subjects meet the following glycemic criteria:

- 1. More than 3 consecutive, daily, fasting SMBG measures are ≥ 270 mg/dL (15 mmol/L) from baseline to week 6, ≥ 240 mg/dL (13.3 mmol/L) after week 6 to week 12, or ≥ 200 mg/dL (11.1 mmol/L) after week 12 to week 96
- 2. Fasting SMBG values are ≥ 250 mg/dL (13.9 mmol/L) and associated with clinical signs or symptoms of hyperglycemia (*e.g.*, weight loss, blurred vision, increased thirst, or increased urination, or fatigue), and the signs or symptoms are severe

From week 0 to week 6, up-titrating glimepiride dose to next higher level should be considered prior to prescribing rescue medication for hyperglycemia. If necessary, increases in glimepiride dosing can occur before the scheduled study visits. The criteria for glimepiride up-titration are provided in Section 3.3.2.1. After glimepiride up-titration to the maximal level, rescue medication should be initiated for treating hyperglycemia based on investigator's assessment.

After week 6 of treatment, no further increases in glimepiride will occur. Therefore, from weeks 7 to 96, rescue medication for hyperglycemia should be prescribed by the investigator when deemed necessary for the well-being of the subject.

If a rescue medication for hyperglycemia is to be prescribed, a blood sample must be drawn prior to the administration of the rescue medication so that a final HbA1c value can be ascribed to the latest date upon which the subject's glycemic control will be impacted by the rescue medication.

The investigator may provide rescue treatment with any approved medication for diabetes that is not otherwise contraindicated, with the exception of SGLT2 inhibitor, sulfonylurea


and metformin, as all study subjects will already be taking metformin and may be taking active SGLT2 inhibitor or glimepiride through study participation.

If hypoglycemia occurs in any subject who has been prescribed rescue medication for hyperglycemia during the study, the total daily dose of the rescue medication should be reduced 50% or more at the discretion of the investigator. If recurrent symptomatic hypoglycemia occurs after discontinuation of the rescue medication or in subjects who are not prescribed rescue medication, study drug can be discontinued at the discretion of the investigator.

Subjects who receive rescue medication due to poor glycemic control will continue to receive investigational products and standard of care per investigator decision, according to current treatment guidelines. Following the exit visit, subjects will be advised to see their primary physician to undergo treatment to control their diabetes.

## 3.3.4 Other Safety Monitoring Activities

The safety monitoring activities will include assessments of vital signs, 12-lead ECG, physical examinations, urinalysis, blood chemistry, hematology, adverse events, and concomitant medication use. The occurrence of blood, liver, or skin disorders will be monitored through laboratory testing and evaluation of adverse event documentation.

Adverse events of special interest as defined in the statistical analysis plan will include any clinical signs and symptoms that indicate adverse experience in the categories listed below. All such events must be appropriately documented within source documentation.

- Genital mycotic infection
- Urinary tract infections including urosepsis and pyelonephritis
- Acid-base disorders including diabetic ketoacidosis
- Diuretic effects including hypovolemia
- Hypotension episodes
- Hepatotoxicity
- MACE
- Hypoglycemia
- Falls and fractures
- Malignancies
- Hypersensitivity reactions
- · Renal failure events
- Amputation

# 3.3.5 Data and Safety Monitoring Board (DSMB)

An independent Data and Safety Monitoring Board (DSMB) will monitor overall safety information during the bexagliflozin development program. The safety review activity and potential risk benefit assessments utilized by the DSMB will be defined in its charter.


### 3.3.6 Major Adverse Cardiovascular Event (MACE) Adjudication

An independent cardiovascular adjudication committee has been established to review, under blind, all potential cardiovascular events occurring during the study. The events of interest include cardiovascular mortality, myocardial infarction (MI), stroke, hospitalization for acute coronary syndromes, urgent revascularization procedures, and other possible serious cardiovascular events. The adjudicated events will be documented and archived to allow a meta-analysis to be performed at a later time. No separate cardiovascular risk assessment will be performed based on events in the study population of the current protocol.

### 3.3.7 Diabetic Ketoacidosis (DKA) Event Adjudication

An independent adjudication committee will be established to review all potential diabetic ketoacidosis events under blind. The adjudicated events will be documented and archived. All adjudicated DKA events in the bexagliflozin phase 3 program will be pooled at the end of the program and a final analysis will be conducted.

## 3.4 Study Duration and Dates

Subjects will be screened within 3 weeks of enrollment. Eligible subjects who provide written consent will start a wash-out and run-in period of 2 or 8 weeks prior to randomization to receive study drugs. Subjects will receive 2 weeks of run-in medication and 96 weeks of treatment and will be followed for 2 weeks after the last dosing. The study duration from screening to follow-up will be no more than 109 weeks overall. For details of the schedule and nature of the investigations, see the Schedule of Events in Appendices 1 and 2.


### 4 STUDY POPULATION SELECTION

# 4.1 Study Population

The study population will include approximately 420 subjects whose T2DM is inadequately controlled by metformin and who meet all of the inclusion criteria, none of the exclusion criteria. Clinical sites in the North America and Europe are anticipated to recruit subjects. Clinical sites in other continents may also participate in the trial.

#### 4.2 Inclusion Criteria

Prospective subjects must be:

- 1. Male or female adult subjects  $\geq$  18 years of age
- 2. If subjects are female of childbearing potential, subjects must be negative on the urine pregnancy test and agree to abstain from coitus or use contraception during the entire study to avoid any possible pregnancy.
- 3. Subjects who are in one of the two categories:
  - a) Metformin-only treated: receive ≥ 1500 mg/day metformin only for at least 8 weeks prior to screening or
  - b) Metformin-and-OHA treated: receive ≥ 1500 mg/day metformin for at least 8 weeks prior to screening and ≥ 14 days of 1 additional oral hypoglycemia agent (OHA) in the 8 weeks prior to screening.
- 4. Subjects with a diagnosis of T2DM with HbA1c levels between 7.0% and 10.5% (inclusive) at screening if metformin-only treated or with HbA1c levels between 6.5% and 10.0% (inclusive) at screening if metformin-and-OHA treated
- 5. Subjects have a body mass index (BMI)  $\leq$  45 kg/m<sup>2</sup> at screening
- 6. If applicable, taking stable doses of treatment for dyslipidemia and/or hypertension for 30 days prior to screening. Subjects do not need to be treated with dyslipidemia or hypertension to be eligible for the study.
- 7. Subjects who are willing and able to return for all clinic visits and to complete all study-required procedures, including self-monitoring blood glucose (SMBG) measurements

Prior to randomization, all subjects must:

- 8. Maintain adequate glycemic control during the washout and run-in periods (fasting plasma glucose values are not  $\geq 250 \text{ mg/dL}$  on consecutive days)
- 9. Have an HbA1c between 7.0% and 10.5% (inclusive) at Visit V5
- 10. Adhere to the investigational product administration requirements as evidenced by missing no more than 2 doses of run-in medications


#### 4.3 Exclusion Criteria

Subjects who exhibit any of the following characteristics will be excluded from the study:

- 1. Diagnosis of type 1 diabetes mellitus or maturity–onset diabetes of the young (MODY)
- 2. Current use of injected therapy for treatment of diabetes (insulin or glucagon-like peptide-1 (GLP-1) receptor agonist therapy) or a thiazolidinedione (TZD)
- 3. Hemoglobinopathy that affects HbA1c measurement
- 4. Any contraindication to the safe use of sulfonylurea therapy, glimepiride or metformin, including known hypersensitivity reaction
- 5. Genitourinary tract infection within 6 weeks of screening or history of  $\geq$  3 genitourinary infections requiring treatment within 6 months from screening
- 6. Cancer, active or in remission, for < 3 years (non-melanoma skin cancer or basal cell carcinoma or carcinoma *in situ* of the cervix will not be grounds for exclusion)
- 7. History of alcohol or illicit drug abuse in the past 2 years
- 8. Evidence of abnormal liver function tests (total bilirubin or alkaline phosphatase > 1.5 x upper limit of normal (ULN) with the exception of isolated Gilbert's syndrome); or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 x ULN
- 9. Estimated glomerular filtration rate (eGFR), as calculated by the modification of diet in renal disease study equation (MDRD), < 60 mL/min/1.73 m<sup>2</sup> at screening.
- 10. Uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure > 95 mmHg) at Visit V1
- 11. History of human immunodeficiency virus (HIV) infection
- 12. Life expectancy < 2 years
- 13. History of myocardial infarction (MI), unstable angina, stroke, or hospitalization for heart failure within 3 months of screening
- 14. History of treatment with an investigational drug within 30 days or within 7 half-lives of the investigational drug, whichever is longer
- 15. Previous treatment with bexagliflozin or EGT0001474 study drug (run-in or double-blind investigational product)
- 16. Currently or within 3 months of taking any SGLT2
- 17. Currently participating in another interventional trial
- 18. Prior renal transplantation or evidence of nephrotic syndrome (defined as a urine albumin-to-creatinine ratio (UACR) > 1500 mg/g at screening).
- 19. Any condition, disease, disorder, or clinically relevant abnormality that, in the opinion of the primary investigator, would jeopardize the subject's appropriate participation in this study or obscure the effects of treatment including condition or co-morbidity for which the use of metformin or any planned or existing second diabetes therapy is contraindicated
- 20. Female subjects who are pregnant or nursing.
- 21. Two or more consecutive SMBG measures ≥ 250 mg/dL (13.9 mmol/L) prior to randomization or severe clinical signs or symptoms of hyperglycemia prior to randomization, including weight loss, blurred vision, increased thirst, or increased urination, or fatigue.


#### 5 STUDY TREATMENTS

# 5.1 Description of Treatments

## 5.1.1 Investigational Product

Bexagliflozin tablets, 20 mg or placebo, are blue caplet-shaped, film-coated tablets that are intended for use in investigational studies in humans. The tablets contain excipients designed to promote extended release through a gastroretentive mechanism. The active tablets exhibit a greater than 75% release of drug substance by 8 h in simulated gastric fluid *in vitro*.

The following investigational products will be used for oral administration:

- Bexagliflozin tablets, 20 mg: tablets containing 20 mg of bexagliflozin
- Bexagliflozin tablets, placebo: tablets containing no bexagliflozin

### 5.1.2 Active Comparator

Glimepiride capsules, 2 mg, 4 mg, 6 mg or placebo, are orange colored capsules.

The following investigational drugs will be used for oral administration:

- Glimepiride capsules, 2 mg: capsules containing 2 mg of glimepiride
- Glimepiride capsules, 4 mg: capsules containing 4 mg of glimepiride
- Glimepiride capsules, 6 mg: capsules containing 6 mg of glimepiride
- Glimepiride capsules, placebo: capsules containing no glimepiride

#### 5.2 Treatments Administered

## 5.2.1 Investigational Product

Bexagliflozin tablets, 20 mg or placebo, should be taken once daily with 250 mL of water in the morning prior to the first meal.

On the day of scheduled clinic visits when there is fasting and blood is to be drawn, administration of bexagliflozin should be delayed until after blood is drawn and taken in the clinic or at home prior to the first meal with 250 mL of water.

## 5.2.2 Active Comparator

Glimepiride is a second generation sulfonylurea, which stimulates glucose-independent insulin release from the pancreas. After oral administration, glimepiride is absorbed from the GI tract. Glimepiride is metabolized mostly by hepatic P450 enzyme CYP2C9.


Glimepiride capsules, 2, 4 or 6 mg or placebo, should be taken once daily with the first meal. On the day of scheduled clinic visits when there is fasting and blood is to be drawn, administration of glimepiride shall be withheld until the first meal.

### 5.2.3 Background Metformin Therapy

Metformin is commonly prescribed as the first-line agent for treating T2DM. It is a biguanide that decreases hepatic glucose production and may improve peripheral glucose uptake and utilization. After oral administration, metformin is absorbed from the gastrointestinal (GI) tract, and it is excreted unchanged in the urine and does not undergo hepatic metabolism or biliary excretion.

Any OHA other than metformin taken by study subjects prior to screening will be discontinued at the start of the wash-out period. Subjects will continue receiving metformin as background therapy during the entire study period at an unchanged dose ( $\geq 1500$  mg/day), time, and frequency that is prescribed to subjects prior to screening.

The dose, frequency, and time of administration should remain stable unless the investigator deems adjustment (decrease or increase) necessary for the medical well-being of the subject. Changes to the dose, frequency, or time of administration of metformin should be recorded in the concomitant medication log.

### 5.2.4 Diuretics and Medications for Treatment of Dyslipidemia and Hypertension

Subjects who are prescribed diuretics, anti-hypertensive agents, or medications to treat dyslipidemia medications to treat hypertension or dyslipidemia will continue the current dose, frequency, and time of administration of these medications throughout the study. Adjustment of these medications will not be permitted during the screening, washout and run-in periods.

If a change in diuretics, anti-hypertensive agents, or medications to treat dyslipidemia is required during the screening or wash-out period, the subject will discontinue study activities and may be re-screened after the clinical condition and treatment regimen have been stable for at least 30 days.

Subjects who start the run-in period or screen fail for any reason, including adjustment of diuretics, anti-hypertensive agents, or medications to treat dyslipidemia, will not be allowed for re-screening.

If a subject re-enters screening after treatment adjustment, a new subject number will be assigned. During the treatment period, adjustments in the treatment for hypertension or dyslipidemia are permitted if required for the well-being of the subject. If it is medically necessary to alter blood pressure medications during the treatment period, new diuretic medications should not be initiated and the dose and frequency of existing diuretic medications should not be changed during the first 2 weeks of therapy. Changes to the dose or frequency of anti-hypertensive and diuretic medications will be recorded in the concomitant medications log.


# 5.3 Selection and Timing of Dose for Each Patient

# 5.3.1 Bexagliflozin

Dosing with bexagliflozin tablets, 20 mg or placebo, will be based on randomized assignment. All study subjects will be instructed to take bexagliflozin tablets once daily in the morning prior to the first meal; bexagliflozin tablets should be taken once daily P.O. with 250 mL water. There will be no change of dose and frequency during the 96-week treatment period.

On the day of each scheduled clinic visit, subjects must fast for approximately 10 h prior to the collection of blood samples. During the fasting period, only water will be permitted.

## 5.3.2 Glimepiride

Dosing with glimepiride capsules or placebo, will be based on randomized assignment at the beginning of the treatment period. The dose of glimepiride may be increased during the first 6 weeks of treatment according to the protocol-specific criteria (Section 3.3.2.1). From weeks 7 to 96, subjects will continue receiving glimepiride at the dose prescribed to them at week 6. Down titration of glimepiride will not be permitted during the entire study period.

# 5.4 Method of Assigning Treatment Groups and Study Drugs

The study will be conducted at multiple investigative sites and will likely involve variable numbers of subjects at each site. Enrollment will be on a competitive basis, but each site will be capped at 40 randomized subjects. Activation of investigational sites in each country will be centrally controlled by an Interactive Web Response System (IWRS).

Eligible subjects who complete the wash-out and run-in period and meet all study inclusion/exclusion requirements will be randomized in a 1:1 ratio to receive active bexagliflozin with placebo glimepiride or active glimepiride with placebo bexagliflozin. Subjects will be assigned to treatment groups in sequential order as they qualify for the study. Randomization will be stratified according to baseline (Visit V5) HbA1c (< 8.5% or  $\ge 8.5\%$ ), treatment background (metformin-only or metformin-and-OHA), and Visit V5 eGFR ( $\ge 90$  or < 90 and  $\ge 60$  mL/min/1.73 m<sup>2</sup>).

The investigator or designated staff will log in to the IWRS to receive the following information:


| Table 2. Study Drug Dispensation Schedul |
|------------------------------------------|
|------------------------------------------|

| Visit | Unique ID | Run-in Drugs | Bexagliflozin Tablets<br>(no. of kits) | Glimepiride Capsules (no.<br>of kits) |
|---|---|---|---|---|
| V1 | Subject no. | | | |
| V4 | | bexagliflozin & glimepiride | | |
| V6 | Randomization no. | | 20 mg or placebo (1) | 2 mg or placebo (1) |
| V7 to V9 <sup>1</sup> | | | | 4 mg, 6 mg or placebo (1) |
| V10 to V14 | | | 20 mg or placebo (1) | 2, 4 or 6 mg or placebo<br>assigned at Week 6 (1) |
| V15 | | | 20 mg or placebo (2) | 2, 4 or 6 mg or placebo<br>assigned at Week 6 (2) |

The investigator will select the glimepiride dose based on clinical assessment. The up-titration of glimepiride dosing can occur before the scheduled study visits in the case of persistent hyperglycemia. The guidance for glimepiride up-titration is outlined in Section 3.3.2.1.

Subject randomization will be deactivated for all sites when the planned number of subjects is met. However, if a potential subject is in wash-out already and wishes to continue with the study, the subject will be allowed to continue and, if eligible, to be randomized.

# 5.5 Blinding

This is a double-blind, double dummy study. The sponsor, investigators, study coordinators, pharmacists, study subjects, the cardiovascular adjudication committee and the diabetic ketoacidosis committee will be blinded to the study medication.

To maintain blinding of the individual treatment assignment, the results of urinary glucose testing will <u>not</u> be made available to any study personnel or subjects. If knowledge of the test substance is needed to manage a subject's condition, the investigator will contact the IWRS to obtain the treatment assignment. If unblinding occurs for any reason, the time and reason for breaking the blind will be recorded on the case report form (CRF) and the sponsor must be notified within 24 h.

A designated statistician who is not involved with the study operation will hold the treatment codes. The unblinded treatment information can be provided to the DSMB to facilitate the evaluation of any clinically important increase in the rate of a serious suspected adverse reaction or to the designated safety contact when the treatment information is required to determine if an expedited safety report must be submitted to regulatory agencies.

The treatment assignment will continue to be withheld from the cardiovascular adjudication committee and diabetic ketoacidosis adjudication committee members until all global investigational studies are completed and final analyses to assess cardiovascular and ketoacidosis risks are conducted.


# 5.6 Concomitant Therapy

During the course of the study, investigators will manage glucose, blood pressure and lipid levels according to local or regional standard of care guidance documents for the management of T2DM. Instructions for intensification of medical therapy for hyperglycemia are provided in Section 3.3.3.3. Instructions and requirements for adjustment to diuretics and treatment for dyslipidemia and hypertension are provided in Section 5.2.4. Subjects will be allowed to take medications or medicinal supplements prescribed to manage non-diabetic medical conditions during the study. Any concurrent medication or supplemental treatment of other, non-diabetes, medical conditions should be continued at a stable dose and frequency for the entire study duration unless there is a clinical reason to change the dose or frequency.

Subjects may receive any medications for adverse events that are necessary in the investigators' judgment. Concomitant medications prescribed at the time of the wash-out and run-in period and during the study are to be recorded on the CRF. The medication name, dose, frequency, route of administration, date(s) of administration and reason for administration must be recorded. This documentation should continue through the treatment period and the follow-up period.

Any medication prescribed to a subject after enrollment and prior to randomization, including contraceptives, must be recorded in the CRF.

#### 5.7 Restrictions

# 5.7.1 Prior Therapy

All subjects will continue regimens for medical conditions other than diabetes during the study as indicated above. No subject shall have been treated with an investigational drug within 30 days of screening or within a period equal to less than 7 half-lives of the investigational drug, whichever is longer. No subject shall have been treated with an SGLT2 inhibitor within 3 months of screening. Subjects taking insulin or GLP-1 receptor agonists or a TZD at the time of screening are not eligible for this study.

#### 5.7.2 Fluid and Food Intake

During the study, subjects will be counseled to remain adequately hydrated at all times. In addition, subjects will receive counseling regarding an appropriate diet to achieve glycemic control based on standards of medical care in diabetes. For example, the recommended diet might be low in saturated fat, high in fiber, and low in simple carbohydrates and contain appropriate caloric intake to maintain weight.

Subjects will fast for approximately 10 h prior to the scheduled blood sample draws. During fasting, only water will be permitted.

#### 5.7.3 Subject Activity Restrictions

Throughout the study period, subjects are counseled and encouraged to engage in a level of physical activity that is appropriate for their physical condition. For those without specific restrictions or limitations, at least 150 min/week of moderate activity is advised by the American Diabetes Association (ADA) (American Diabetes, 2014). Alternatively, local regulatory guidelines may be used.

#### 5.8 Treatment Compliance

Subjects will be provided with dosing instructions when the investigational products are dispensed. Subjects will also be instructed to bring their medications with them at every visit. During the run-in period, subjects will be excluded from randomization if more than 2 placebo run-in medication doses of any kind have been omitted.

At each visit the study staff will review SMBG diary and medications use with the subject and record the drug consumption in the CRF. Reasons for non-adherence will also be recorded in the protocol deviation log if applicable.

#### 5.9 Packaging and Labeling

Investigational products will be provided to the pharmacist or designated site personnel in high-density polyethylene (HDPE) bottles of 90 tablets enclosed with a child-resistant cap. A bottle of 15 bexagliflozin tablets, placebo, and a bottle of 15 glimepiride capsules, placebo, will be provided for the 2-week run-in portion of the study. All investigational product supplies will be prepared and labeled according to the requirements of local laws and regulations. The pharmacist or designated site personnel will dispense the investigational products for each subject according to randomization assignment.

#### 5.9.1 Run-in Kits

Two types of run-in kits are provided:

- Bexagliflozin tablets, placebo, 15 tablets per bottle;
- Glimepiride capsules, placebo, 15 capsules per bottle.

The label attached to each run-in kit will contain the protocol number, product identification, kit number, batch number, expiration date, subject number, investigator name, storage condition, directions for use, sponsor's name and address, and the investigational drug caution statement.

#### 5.9.2 Bexagliflozin Kit

One bexagliflozin kit contains a bottle of 90 counts of bexagliflozin tablets, 20 mg or placebo.


The label attached to each bexagliflozin kit will contain the protocol number, product identification, kit number, batch number, expiration date, subject number, investigator name, storage condition, directions for use, sponsor's name and address, and the investigational drug caution statement.

#### 5.9.3 Glimepiride Kit

One glimepiride kit contains a 90 count bottle of one of the following products:

- Glimepiride capsules, 2 mg or placebo
- Glimepiride capsules, 4 mg or placebo
- Glimepiride capsules, 6 mg or placebo

The label attached to each glimepiride kit will contain the protocol number, product identification, kit number, batch number, expiration date, subject number, investigator name, storage condition, directions for use, sponsor's name and address, and the investigational drug caution statement.

#### 5.10 Storage and Accountability

Bexagliflozin tablets and glimepiride capsules will be stored at controlled room temperatures of 15°C to 30°C (59°F to 86°F). The sponsor will notify the sites of the process for returning unused drug.

### 5.11 Investigational Product Retention at Study Site

The investigational products will be stored in a secure area with limited access. The drug storage facility must comply with the medication storage instructions. The investigational products should be stored at controlled room temperature until ready for dispensing to study subjects. The trial staff must record the amount of investigational products dispensed to each subject on the dosing record. To ensure adequate recordkeeping, subjects must bring all investigational products to each visit. The remaining tablets and capsules will be accounted for in the CRF and drug consumption forms. The procedures for obtaining drug resupply will be provided by the sponsor. All unused drug must be returned to a sponsor-designated depot after drug accountability is verified by the sponsor or its designee.


#### 6 STUDY PROCEDURES

#### 6.1 Informed Consent

Before each subject is enrolled in the clinical study, written informed consent will be obtained according to the regulatory and legal requirements of the participating country. As part of this procedure, the investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study subject is aware of the potential risks, inconveniences, or adverse events (AEs) that may occur. The investigator should educate potential subjects about the scientific importance of their data and the vital role that their participation has for the outcome of the entire study. The subject must be informed that he/she is free to withdraw from the study at any time. He or she will receive all information that is required by federal regulations and International Council for Harmonisation (ICH) guidelines.

The informed consent document must be signed and dated; one copy will be given to the patient, and the investigator will retain a copy as part of the clinical study records. The investigator will not undertake any investigation specifically required for the clinical study until written consent has been obtained. The terms of the consent and when it was obtained must also be documented

#### 6.2 Screening for I/E Criteria

At the initial screening, the investigator should review the inclusion and exclusion criteria based on the information collected at the screening visit. Any change to status affecting conformance to inclusion and exclusion criteria at subsequent visits prior to randomization must be evaluated. At randomization, the investigator should confirm the run-in drug compliance.

## 6.3 Medical History

The following information will be collected at the screening visit:

### 6.3.1 General Demographics and Characteristics

- 1. Date of birth, age, sex, and race, and whether a female subject is of childbearing potential or not.
- 2. Significant medical and surgical history, including dates of diagnoses and procedures and whether the condition is ongoing, if applicable.

#### 6.3.2 Diabetes History

1. History of all medications used to treat diabetes (to be recorded in the concomitant medication form), including start date, duration of use, and stop date, if applicable.


- 2. History of complications due to diabetes, including nephropathy, retinopathy, neuropathy, non-traumatic amputations, and diabetic ketoacidosis, including date of diagnosis
- 3. Frequency of hypoglycemic events (per week) that are symptomatic or require assistance.

#### 6.3.3 Cardiovascular Disease History

History of cardiovascular disease including presence of angina, congestive heart failure (including New York Heart Association [NYHA] classification), known atherosclerotic cardiovascular disease, prior MI, transient ischemic attack or stroke, and prior cardiac or peripheral re-vascularization procedures. The history should include the date of diagnosis and the current status of diagnosis (resolved or ongoing).

#### 6.3.4 Medication History

- 1. Use of prescribed or non-prescribed medications, including name of medication, indications for usage, start and stop dates, dose, and frequency
- 2. Use of supplements, including over the counter drugs, vitamins, herbal preparations, and dietary supplements within the past 30 days prior to screening. Each medication history will include the agent used, indication for usage, start and stop dates, dose, and frequency.

#### 6.4 Diet and Exercise Counseling

Subjects will receive counseling regarding an appropriate diet and exercise regimen to aid in glycemic control based on standards of medical care in diabetes throughout the study. In addition, all subjects are encouraged to consume enough liquid to maintain adequate hydration.

## 6.5 Physical Examination

A complete physical examination will be performed by the investigator at the time points indicated in the Schedule of Events (Appendix 1). The examination will include measurement of body weight and height (height will be measured only at screening), general assessment of all body systems including the skin, head, eyes, ears, nose, throat, neck, heart, lungs, abdomen, lymph nodes, and extremities.

The body weight must be determined using a scale that is calibrated. The same scale should be used throughout the study duration.

## 6.6 Abbreviated Physical Examination

An abbreviated physical examination will include body weight and general assessment of the skin, heart, lungs and abdomen. Abbreviated physical examinations will be performed by the investigator at the time points indicated in the Schedule of Events (Appendix 1), unless clinically indicated.


The body weight must be determined using a scale that is calibrated. The same scale should be used throughout the study duration.

#### 6.7 Vital Signs

Vital signs will be measured at the time points indicated in the Schedule of Events (Appendix 1) and will include supine, sitting and standing BP measurements, and heart rate.

Devices designed to measure BP from the finger or wrist may not be used. The left arm and same cuff sizes should be used for each measurement at all visits. If the left arm cannot be used at the screening visit or during the study for BP measurements, the reason should be documented, and the right arm should be used for BP measurements for all subsequent visits.

At each visit, BP measurements will be obtained using a calibrated sphygmomanometer while the subject is in sitting, supine, and standing positions. A single heart rate measurement should be taken just prior to the BP evaluation in the sitting, supine, and standing positions.

All readings are to be entered into the source document and CRF for all subjects. The date and time of BP measurements should be captured in the source document and CRF. BP will be assessed first in the sitting position. Sitting BP and heart rate will be measured after the subject has been sitting for at least 5 minutes with feet on the floor and arm supported at heart level.

After sitting BP measurement has been completed, supine and standing BP will be measured to evaluate orthostatic vital signs. Supine and standing blood pressure measures will not be used to determine eligibility for the study. First, the subject will lie flat for 5 minutes and have heart rate and supine blood pressure measured using the same equipment and arm as described for sitting BP. Once the supine BP measurement is complete, the subject will stand. Standing BP and heart rate will be measured after 2 minutes of standing. For standing BP measurements, the arm should be supported and extended such that the cuff is at heart level

## 6.8 Electrocardiography

A 12-ECG will be conducted at the time points indicated in the Schedule of Events in Appendix 1 and whenever clinically indicated. This procedure should be performed in the supine position after at least 10 min of rest. ECG parameters measured will be the RR interval, PR interval, QRS duration, and QT interval. Each ECG should also be assessed by the investigator for signs of ischemia, clinically significant hypertrophy, and clinically significant T-wave abnormalities or arrhythmia.

It is the investigator's responsibility to review the results of the ECG as they become available. For each abnormal ECG result, the investigator shall ascertain if the observation represents a clinically significant change from the screening ECG for that individual subject. This determination does not necessarily need to be made the first time an abnormal result is observed. The investigator may repeat the ECG to verify the original result. If the ECG result


is determined to be a clinically significant and abnormal change from baseline for that subject, it is considered to reflect an AE.

#### 6.9 Clinical Laboratory Tests

#### 6.9.1 Laboratory Parameters

Clinical laboratory tests are listed in Table 3.

- 6.9.2 Sample Collection, Storage, and Shipping
- 6.9.2.1 Hematology, Blood Chemistry, Serum Lipids, and Glycemic Control Assessments

Blood samples for hematology, chemistry, serum lipids and glycemic control assessments will be collected. Subjects will be in a seated or supine position during blood collection. Samples will be collected at the time points indicated in the schedule of events in Appendix 1 and Appendix 2.

The study staff will contact each subject prior to a scheduled clinic visit to confirm the time of the visit and to remind the subject of proper fasting practice. A subject must be queried to assess compliance with an approximately 10 h fast prior to blood draw to ensure the FPG and triglycerides values can be accurately determined. If a subject has not fasted for approximately 10 h, the subject must return as soon as can be arranged (within 1 week) to provide a specimen after proper fasting.

Low-density lipoprotein-cholesterol (LDL-C) will be calculated by the Friedewald equation. If triglycerides are > 400 mg/dL, the calculated LDL-C value is invalid by this equation and will be set as missing. Direct LDL-C will be determined in subjects whose triglycerides are > 350 mg/dL at screening visit. All subsequent LDL-C of these subjects will be determined by the same direct LDL-C measurements only.

#### 6.9.2.2 Urinalysis

Urine samples will be collected routinely at designated clinic visits from a clean catch sample. Urinalysis will be performed at the time points indicated in the schedule of events (Appendix 1 and Appendix 2). Investigator or staff should document if pre-menopausal female subjects are menstruating and note it in the source documents since hematuria is likely to be identified on dipstick urinalysis.

Urine samples will be transported to the central laboratory for urinalysis. Microscopy will be conducted if the subject has a positive result on the leukocyte esterase or nitrite dipstick tests to clarify the significance of the finding. Results of glucose measurement in the urinalysis must be suppressed from the laboratory reports so the sponsor, investigators, study coordinators, pharmacists, study subjects, the cardiovascular endpoint committee (CEC) members and (diabetic ketoacidosis) DKA adjudication committee members will remain blinded to the dosing assignment.


In addition, strips to assess leukocyte esterase and nitrite but not glucose will be provided for immediate assessment at the clinical sites. If more than traces of positive results are shown in the leukocyte esterase and /or nitrite testing, a urine culture should be performed in a designated laboratory regardless of patient reported signs or symptoms. Results of the urinalysis and possible urine culture will be documented in the CRFs.

Renal functional testing by UACR will be determined at time points specified in the schedule of events (Appendix 1 and Appendix 2).

#### 6.9.2.3 Urine Pregnancy Test (UPT)

UPT will be performed for all women, including surgically sterile or post-menopausal women, at the screening visit. Additionally, women of child bearing potential (WOCBP) will receive a UPT at the clinical visits indicated in Appendix 2.


Table 3. **List of Laboratory Tests** Test Name (sample volume) Hematology (2 mL blood) • Mean corpuscular hemoglobin • Mean corpuscular volume (MCV) • Red blood cell (RBC) count (MCH) • White blood cell (WBC) count • Hematocrit (Hct) with differential • Mean corpuscular hemoglobin Hemoglobin (Hgb) concentration (MCHC) RBC Morphology · Platelet count Serum Chemistry and Electrolytes (3 mL serum) • Albumin (ALB) • Calcium (Ca) Glucose ALT Magnesium • Bicarbonate (HCO<sub>3</sub>) Phosphorus AST • Chloride (Cl) • Blood urea nitrogen (BUN) • Potassium (K) Total bilirubin Creatinine • Sodium (Na) Direct bilirubin • Uric acid • Total Protein Glycemic Control (2 mL plasma, 2 mL blood) • FPG • HbA1c Serum Lipids Triglycerides (TG) • Total cholesterol (TC) • Low-density lipoprotein cholesterol (LDL-C), calculated, • High-density lipoprotein cholesterol (HDL-C) • LDL-C, direct (if applicable) Urinalysis Appearance • Microscopic examination of • pH sediment Bilirubin Protein • Nitrite Color Specific gravity • Leukocyte esterase • Glucose (blinded) • Urobilinogen · Occult blood Ketones Renal Functional Test UACR

## 6.10 Diary and Glucometer Dispensation and Review

**Urine Pregnancy Test** 

A glucometer, testing strips, and a glycemic control diary will be provided to each metformin-and-OHA treated subject at the start of wash-out and each metformin-only treated subject at the start of run-in. Subjects will be trained to use the glucometer and record any events in the glycemic control diary. Study subjects may continue using their own glucometer, if applicable, if the device has a function for glucose value storage for at least 180 days and the glucose values must be downloadable so that SMGB records can be kept for


the evaluation by the investigator. The SMBG record from the glucometer and diary entries must be reviewed by the investigator at all subsequent visits including both phone interview and clinic visits.

During the SMBG training, symptoms that may indicate hypoglycemia, hyperglycemia, or ketoacidosis will be reviewed with study subjects. Instructions to contact the clinic when the subjects experience potential hypoglycemia or diabetic ketoacidosis must be provided.

#### 6.11 Dispensing Run-in Drug

Each eligible study subject will receive 1 bottle of bexagliflozin, placebo run-in drug and 1 bottle of glimepiride, placebo run-in drug based on the scheduled visit outlined in Appendix 1.

#### 6.12 Diary and Glucometer Record Review

Review SMBG and glycemic control record.

#### 6.13 Dispensing Investigational Product

#### 6.13.1 Dispensing Bexagliflozin

At randomization and at every 12 weeks of treatment thereafter, each study subject will receive 1 bottle of bexagliflozin tablets, 20 mg or placebo, based on the kit number assigned to the subject by the IWRS. At visit V15, two bottles of bexagliflozin tablets will be dispensed for dosing between week 72 and week 96.

#### 6.13.2 Dispensing Glimepiride

#### Weeks 0 to 6

- Each subject will receive 1 bottle of glimepiride capsules, 2 mg or placebo, at randomization.
- During weeks 2 to 6 post-randomization, the investigator will select the glimepiride dose based on clinical assessment. The guidance for glimepiride up-titration is outlined in Section 3.3.2.1. If subjects meet up-titration criteria, a bottle of glimepiride, 4 mg, 6 mg or placebo, will be dispensed. If subjects do not meet up-titration criteria, subjects will continue the glimepiride prescribed to them at the previous visit. The up-titration of glimepiride dosing can occur before the scheduled study visits in the case of persistent hyperglycemia.

#### Weeks 7 to 96

- From weeks 7 to 12, each subject will continue taking glimepiride prescribed to them at week 6.
- At week 12 and at every 12 weeks of treatment thereafter, each study subject will receive 1 bottle of glimepiride capsules, 2mg, 4 mg, 6 mg or placebo, based on the kit number


assigned to the subject by the IWRS. At visit V15, two bottles of glimepiride capsules will be dispensed for dosing between week 72 and week 96.

#### **6.14 Adverse Events Assessments**

#### 6.14.1 Definition of Adverse Events

**Adverse event (AE):** Any untoward medical occurrence in a subject administered a pharmaceutical product that does not necessarily have a causal relationship with the treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not it is considered related to the medicinal product use.

**Serious adverse event (SAE):** A serious adverse event (experience) or reaction is any untoward medical occurrence that at any dose:

- 1. results in death,
- 2. is life-threatening, (NOTE: The term "life-threatening" in this context refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe.)
- 3. requires inpatient hospitalization or prolongation of existing hospitalization,
- 4. results in persistent or significant disability/incapacity,
- 5. is a congenital anomaly/birth defect, or
- 6. is a medically important event or reaction. Medical and scientific judgment should be exercised in deciding whether other situations should be considered serious such as important medical events that might not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes listed in the definition above. These should also usually be considered serious. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

**Adverse Reaction:** An adverse reaction means any adverse event caused by a drug. Adverse reactions are a subset of all suspected adverse events in which there is a reason to conclude that the drug caused the event.

**Unexpected Adverse Drug Reaction (UADR):** An adverse reaction, the nature or severity of which is not consistent with the applicable product information (see the Investigator's Brochure for an unapproved investigational medicinal product).

**Serious and Unexpected Suspected Adverse Reaction (SUSAR):** The sponsor must report in an Investigational New Drug (IND) safety report any suspected adverse reaction to study treatment (including active comparators) that is both serious and unexpected (21 CFR


312.32(c)(1)(i)). Before submitting an IND safety report, the sponsor needs to ensure that the event meets all three of the definitions:

- Suspected adverse reaction
- Serious
- Unexpected

**Severity:** AEs will be graded on a 3-point scale and reported as indicated in the CRF. The intensity of an adverse experience is defined as follows:

- 1 = Mild: event is medically significant but produces no disruption to daily activity;
- 2 = Moderate: event is medically significant and reduces or affects normal daily activity;
- 3 = Severe: event is medically significant and results in inability to work or perform normal daily activity.

**Investigational Product Causality:** An assignment will be made by the investigator based on the circumstances of the event and its analysis. Cases with causal relationship classified as possible, probable or definite are defined as related. Cases with causal relationship categorized as not likely or unrelated are defined as not related. Relationship of an AE to dosing will be assessed as follows:

**Definite:** The event responds to withdrawal of the investigational product (dechallenge), and recurs with rechallenge by administration of the investigational product.

**Probable:** There is a reasonable causal relationship between the investigational product and the AE. The event responds to dechallenge. Rechallenge is not required.

**Possible:** There is a reasonable causal relationship between the investigational product and the AE. Dechallenge is lacking or dechallenge response is unclear.

**Not Likely**: There is a temporal relationship to investigational product administration, but there is not a reasonable causal relationship between the investigational product and the event.

**Unrelated:** There is not a temporal or causal relationship to investigational product administration.

#### 6.14.2 Eliciting and Reporting AEs

The investigator will periodically assess each subject for the occurrence of AEs after the subject consents to participation in the study. To avoid bias in collecting information about AEs, the investigator should ask subjects the following question: "How have you felt since you were last checked?" All AEs (serious and non-serious) reported by the subject must be recorded on the source documents and CRFs provided by the sponsor.


It is the investigators responsibility to review the results of all laboratory tests as they become available. For each abnormal laboratory test result the investigator needs to ascertain if the result is a clinically significant change from baseline for that individual subject. This determination, however, does not necessarily need to be made the first time an abnormal value is observed. The investigator may repeat the laboratory test or request additional tests to verify the results of the original laboratory tests. If the laboratory value is determined to be a clinically significant and an abnormal change from baseline for that subject, the result is considered a laboratory AE.

Hypoglycemia is defined as any FPG or SMBG value  $\leq 70$  mg/dL and documented as described in Section 6.14.11.

Any increase in liver function tests (AST, ALT, or bilirubin) greater than 3 times the ULN for the laboratory utilized will automatically be considered a laboratory AE unless the investigator specifically designates otherwise. In addition, investigators are reminded that any increase in liver function test values that fall below this threshold may be considered clinically significant and entered as an AE if the change is determined to be clinically significant.

In addition, the sponsor's Medical Monitor or its designated personnel must be notified immediately by telephone, email, or fax of any immediately reportable AEs (IRAE) according to the procedure outlined below. Special attention should be paid to recording hospitalization and concomitant medications.

#### 6.14.3 Immediately Reportable AEs

The investigator must report any SAE to the sponsor or its representative immediately after the investigator becomes aware of the event. An SAE form should be completed and sent to the sponsor or representative within 24 h of knowledge of the event.

Non-serious events that require discontinuation of investigational product (including laboratory abnormalities) should be reported to the sponsor within 3 working days. The CRF AE form should be completed and sent to the sponsor.

Subjects experiencing an SAE should be followed clinically until their health has returned to baseline status or no further improvement in condition can be expected with further care. It is expected that the investigator will provide or arrange appropriate supportive care for the subject.

#### 6.14.4 Pregnancy

WOCBP who are sexually active must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized.

Before enrolling WOCBP in this clinical trial, investigators must review guidelines about study participation for WOCBP. The topics should generally include:


- General information
- Informed consent form
- Pregnancy prevention information
- Drug interactions with hormonal contraceptives
- Contraceptives in current use
- Guidelines for the follow-up of a reported pregnancy

Prior to study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. The subject must sign an informed consent form stating the above-mentioned risk factors and that the consequences were discussed with her.

During the study, all WOCBP should be instructed to contact the investigator immediately if they suspect they might be pregnant (*e.g.*, missed or late menstrual cycle).

If a subject or investigator suspects that the subject may be pregnant prior to investigational product administration, the investigational product administration must be withheld until the results of serum pregnancy tests are available. If the pregnancy is confirmed, the subject must not receive the investigational product and must not be enrolled or remain in the study. If pregnancy is suspected while the subject is receiving study treatment, the investigational product must be withheld immediately until the result of the pregnancy test is known. If pregnancy is confirmed, the investigational product will be permanently discontinued and the subject will be withdrawn from the trial. (Exceptions to study discontinuation may be considered for life-threatening conditions only after consultations with the sponsor Medical Monitor or designated personnel.) The investigator must notify the Medical Monitor within 3 working days of any female subject who becomes pregnant. This reporting requirement will continue until 4 weeks after the last investigational product exposure.

The investigator must record the event on the Pregnancy Surveillance Form and forward it to sponsor's Medical Monitor or designated personnel.

Protocol-required procedures for study discontinuation and follow-up must be performed on the subject unless contraindicated by pregnancy (*e.g.*, x-ray studies). Other appropriate pregnancy follow-up procedures should be considered if indicated. In addition, the investigator must report to the sponsor, on the appropriate Pregnancy Surveillance Form, follow-up information regarding the course of the pregnancy, including perinatal and neonatal outcome. Infants will be followed for a minimum of six months.

#### 6.14.5 Procedure for Breaking the Blind

As indicated in Section 5.5 above, the sponsor, medical monitor, study coordinators, pharmacists, study subjects, the CEC members and DKA adjudication committee members will be blinded to the treatment assignment during the study period. The investigator should also remain blinded to the subject treatment during the entire study unless knowledge of the subject's treatment is required for clinical care and safety. The Emergency Code Break module in the IWRS is used for such situations. The investigator must confirm the intention to unblind the subject's treatment to obtain the dose information in IWRS. Upon completion


of the unblinding, the system will send an alert to designated study team members that an unblinding event has occurred. Documentation of breaking the blind should be recorded in the subject's medical record with the date and time the blind was broken, and the names of the personnel requesting and authorizing unblinding. The treatment assignment will continue to be withheld from the CEC members.

#### 6.14.6 Follow-up of Non-Serious AEs

Non-serious AEs that are identified on the last scheduled contact must be recorded in the AE CRF with the current status noted. All non-serious events that are ongoing at the time will be recorded as ongoing in the CRF.

#### 6.14.7 Follow-up of Post-Study SAEs

SAEs that are identified on the last scheduled contact must be recorded on the AE CRF page and reported to the sponsor according to the reporting procedures outlined in Section 6.14. These may include unresolved previously reported SAEs, or new SAEs. The investigator should follow these SAEs until the events are resolved, or the subject is lost to follow-up. Resolution means the subject has returned to the baseline state of health, or the investigator does not expect any further improvement or worsening of the subject's condition. The investigator should continue to report any significant follow-up information to the sponsor until the event has been resolved.

Any new SAEs reported by the subject to the investigator that occur after the last scheduled contact, and are determined by the investigator to be reasonably associated with the use of the investigational product, should be reported to the sponsor or designated personnel. This may include SAEs that are captured on follow-up telephone contact or at any other time point after the defined study period (*i.e.*, up to last scheduled contact). The investigator should follow SAEs identified after the last scheduled contact until the events are resolved, or the subject is lost to follow-up. The investigator should continue to report any significant follow-up information to the sponsor until the event has been resolved. This study requires that subjects be actively monitored for SAEs for at least 4 weeks after the last treatment.

#### 6.14.8 Urinary Tract Infections (UTIs)

Events potentially representing UTIs, including cystitis, urethritis, pyelonephritis, or urosepsis, should be carefully evaluated and documentation of signs, symptoms, culture results for infectious agent, and treatment should be undertaken when appropriate.

The investigator should query the subject at every clinical visit for symptoms that may be related to a UTI and, if appropriate, document these events as symptomatic UTI in the CRF unless an alternative diagnosis is present. In addition, a clean catch urine sample will be obtained at all clinical visits and a urinalysis will be performed on that sample at every clinical visit. A positive urinalysis will be defined as one with detectable leukocyte esterase and/or nitrites. If the subject reports symptoms consistent with a UTI or the urinalysis at the clinical site is positive, a urine culture will be performed at the central laboratory. A positive


urine culture will be defined as one with  $\geq 10^5$  CFU of any species. The investigator may also perform a urine culture using local resources if necessary for clinical care.

#### 6.14.9 Genital Mycotic Infections (GMIs)

The investigator will query the subjects for signs or symptoms that may represent a GMI at all clinic visits. GMIs will be diagnosed based on symptoms and, if appropriate, physical exam and laboratory findings. Investigators must exclude the possibility of sexually transmitted infections before diagnosing GMI. Diagnosis of GMIs must be documented in the CRF.

#### 6.14.10 Hepatotoxicity

If plasma AST and/or ALT concentrations > 3 x ULN are detected, the investigator will record in the source documents the date corresponding to the date of the laboratory abnormality, the type, frequency, and dose of any concurrent medications or supplements taken by the subject within the 14 days of the detected abnormality; and any symptoms or change in physical exam that have occurred since the prior assessment. The investigator should perform additional laboratory and imaging tests to attempt to establish the cause of the AST and ALT elevations, including ruling out any potential contribution from bone or muscle etiologies.

Any clinically significant increase in hepatic enzymes and specifically any ALT or AST > 3 x ULN requires immediate repeat test within 48 to 72 h to confirm the hepatic enzyme elevation and should be repeated based on the clinical situation at least every 96 h (4 days) until ALT and AST return to < 2.5 x ULN. Study medication should be stopped and the event should be reported as a laboratory AE within the CRF if the enzyme elevation is confirmed or worsening.

Hepatotoxicity will be diagnosed and entered as an AE should any of the following occur:

- ALT or AST  $> 8 \times ULN$
- ALT or AST > 3 x ULN and total bilirubin > 2 x ULN or INR > 1.5
- ALT or AST > 3 x ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%).

In the event of hepatotoxicity, investigational product should be discontinued. If no alternative cause of hepatotoxicity to the study drug is identified, the study drug should not be restarted. If an alternative cause of hepatotoxicity is identified, study drug administration may be resumed after the liver function testing returns to baseline and any related symptoms have resolved. If the liver function abnormalities or related symptoms recur after dosing is resumed, the study drug dosing should be permanently discontinued. The investigator is encouraged to consult with the Medical Monitor regarding diagnostic evaluation for the hepatic enzyme elevations. Consultation with a hepatologist may also be appropriate in some circumstances.


#### 6.14.11 Hypoglycemia

Events of hypoglycemia or potentially representing hypoglycemia should be carefully evaluated.

All subjects will be provided with a glucometer and diary for recording blood glucose measurements and signs and symptoms of hypoglycemia. During the study the subject is expected to record daily SMBG readings and all signs and symptoms that may potentially reflect hypoglycemia. In the event of such signs or symptoms, the subject is expected to check the blood glucose if it is reasonably safe to do so, and consume carbohydrates, if appropriate, to treat hypoglycemia.

The subject will be expected to record in the glycemic control diary the following information for each hypoglycemic event:

- 1. Signs and symptoms attributed to hypoglycemia and the time and date on which they occurred
- 2. SMBG reading at the time of the signs and symptoms attributed to hypoglycemia
- 3. Time elapsed from the most recent meal to the onset of signs and symptoms
- 4. Duration, intensity, and type of any exercise within the 24 h prior to the signs and symptoms
- 5. Type of treatment used (*e.g.*, juice, crackers) for the signs and symptoms and whether assistance was required from another person to administer the treatment
- 6. SMBG reading 15 minutes after treatment with carbohydrate and the time at which this was measured
- 7. Whether or not the signs and symptoms attributed to hypoglycemia resolved after blood glucose returned to normal.

Subjects are encouraged to call the study clinic should signs and symptoms potentially related to hypoglycemia occur.

At each study visit, the investigator is expected to review the glucometer and glycemic control diary with particular attention to any SMBG value  $\leq 70$  mg/dL and any recorded signs or symptoms potentially related to hypoglycemia. In addition, the investigator should query the subject with regard to the occurrence of signs and symptoms potentially related to hypoglycemia even if none are recorded in the diary.

In the event of a blood glucose value  $\leq 70 \text{ mg/dL}$  or signs and symptoms potentially related to hypoglycemia, the investigator should complete the supplemental CRF which will include data from the glycemic control diary and action items to reduce future hypoglycemia episodes.

Hypoglycemia events will be recorded in the hypoglycemia log under 5 categories:


- 1. Severe hypoglycemia: an event requiring assistance by another person to actively administer carbohydrate, glucagon, or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma. Plasma glucose measurements may not be available during such an event, but neurological recovery attributable to the restoration of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration. All such events should be recorded as SAEs in the CRF.
- 2. Documented symptomatic hypoglycemia: an event during which typical symptoms of hypoglycemia are accompanied by a measured plasma glucose concentration ≤ 70 mg/dL (3.9 mmol/L).
- 3. Asymptomatic hypoglycemia: an event not accompanied by typical symptoms of hypoglycemia but with a measured blood glucose concentration ≤70 mg/dL (3.9 mmol/L).
- 4. Probable symptomatic hypoglycemia: an event during which symptoms of hypoglycemia are not accompanied by a blood glucose determination but that is presumably caused by a blood glucose concentration ≤ 70 mg/dL (3.9 mmol/L).
- 5. Relative hypoglycemia: An event during which the person with diabetes reports any of the typical symptoms of hypoglycemia, and interprets those as indicative of hypoglycemia, but with a measured plasma glucose concentration > 70 mg/dL (3.9 mmol/L).

While each event meeting the criteria above will be entered into the hypoglycemia log, only critical hypoglycemia, documented symptomatic hypoglycemia, asymptomatic hypoglycemia, and probable hypoglycemia will be entered as AEs.

In the event of asymptomatic hypoglycemia, the investigator should review the signs and symptoms of hypoglycemia with the subject to elicit a complete description and should review proper glucometer technique to ensure that the low glucose value is not due to improper use of the glucometer.

The investigator should be alerted to the likelihood of improper glucose measurement technique if a study subject reports an SMBG value < 55 mg/dL that is not associated with any signs or symptoms of hypoglycemia and is not treated by some form of glucose administration.

In the event of probable symptomatic hypoglycemia, the investigator should encourage the subject to obtain glucose values, when possible, in the context of signs and symptoms of hypoglycemia, even if the glucose value is measured after treatment for the symptoms is administered.

If hypoglycemia occurs in any subject prescribed rescue medication for hyperglycemia during the study, the total daily dose of the rescue medication should be reduced 50% or more at the discretion of the investigator.


#### 6.14.12 Diabetic Ketoacidosis (DKA)

DKA is a serious, acute complication of diabetes and can be life-threatening. Subjects will be educated on the signs and symptoms of DKA and are required to call the study clinic and seek treatment should such signs and symptoms occur.

During the clinical trial period, potential DKA will be monitored by the routine measurement of urinary ketones and assessment for signs or symptoms of acidosis at every clinic visit. Clinical presentations, such as difficulty breathing, abdominal pain, nausea, vomiting, lethargy, or a fruity smell in the breath, or laboratory values that suggest clinically significant acidosis should be documented. Treatment of DKA should be provided when appropriate.

If ongoing symptoms or signs suggest a possible DKA, the investigator should perform relevant laboratory testing while directing appropriate medical care for the subject. If DKA is suspected, regardless of the blood glucose level, the following assessments should be done immediately: physical exam and serum glucose, bicarbonate, electrolytes, and serum ketones measured STAT at a local laboratory. If ketoacidosis is likely, investigational product administration should be discontinued and immediate appropriate medical therapy, including insulin, should be initiated. A glucose infusion may be provided if necessary to avoid hypoglycemia during insulin therapy. Insulin treatment should continue until resolution of the ketoacidosis and stabilization of the subject's clinical condition. Investigational product administration may be resumed following stabilization of the subject's condition. Investigator should collect the data necessary for the completion of the DKA CRF.

If symptoms suggestive of DKA may have occurred but are not ongoing, investigator should review available data in order to complete the DKA CRF. The investigator may also perform laboratory assessment using local resources if necessary for clinical care.

#### 6.14.13 Major Adverse Cardiovascular Event (MACE)

Evaluation of MACE will be undertaken across the development program for bexagliflozin. All MACE reports should also be captured as SAEs and every effort will be made to ensure that events recorded as MACE are coded in a similar manner within the safety database. The SAE listing will also be reviewed periodically by the CEC members to identify potential MACE that may not have been reported by the site investigators. All subjects will be followed by investigators for MACE for the duration of the study even if study medication has been permanently withdrawn.

The independent CEC will receive and adjudicate the following events.

- All deaths
- Suspected non-fatal myocardial infarction (MI)
- Suspected hospitalization for unstable angina (HUA)
- Suspected transient ischemic attack (TIA) and stroke
- Suspected hospitalization for heart failure (HF)
- Reported coronary revascularization procedure


#### 6.14.14 Amputation

Amputation and related adverse events will be recorded in a case report form. During each study visit, the investigator should query the subject for any amputation and related adverse events and procedures. Investigators are reminded to counsel appropriate foot care to avoid cuts or sores and to treat even minor cuts or sores to prevent infection and ulceration. Patients who have had a previous amputation should be closely monitored. Special attention may be appropriate for patients who are also receiving thiazide diuretics as these have been shown to increase the risk of amputation in diabetics.

#### 6.15 Concomitant Medication Assessments

A concomitant medication is any medication that the subject has been taking prior to enrollment and that the subject is expected to continue to take for some portion of the trial, as well as any medication other than the investigational product that the subject takes during the course of the trial.

The medications or treatment for controlling hypoglycemia must be recorded as concomitant medications in the CRF. Any medication given to treat hyperglycemia and continued for more than 2 weeks is considered a rescue therapy and should be recorded in the concomitant medication log.

Changes from baseline anti-hypertensive and anti-hyperlipidemia therapies and their rationale must be recorded in the CRF.

All prescription and over-the-counter medications, including vitamins and herbal supplements, that subjects receive during the trial must be documented on the CRF. This documentation should continue until the subjects complete the study.

Concomitant medications will be coded using the World Health Organization Drug Dictionary (WHO-DD). A table of concomitant medications based on the anatomic therapeutic chemical classification (ATC) and preferred name will be produced. A listing of concomitant medications will include all medications taken by any subjects during the course of the study.

## 6.16 Healthy-related Quality of Life Assessment

EQ-5D-3L is a multi-attribute utility instrument for measuring preferences associated with an individual's health state. The instrument includes a visual analog scale and a descriptive system with 5 dimensions (mobility, self-care, usual activity, pain/discomfort, anxiety/depression), each of which has 3 levels (no problem, some problem, extreme problem).

Enrolled subjects will complete the EQ-5D-3L questionnaire independently at clinic Visits V6, V11, V14 and V17. EQ-5D-3L should be completed prior to other scheduled procedures at those visits


# 6.17 Removal of Subjects from the Trial or Discontinuation of Investigational Product Administration

The investigator must emphasize to potential subjects the importance of continued participation for the full duration of the trial during the informed consent process. Potential subjects should be informed that the trial procedures will allow additional medications to control hyperglycemia or other adverse conditions. It is also important to emphasize that missing data and missed visits could affect the entire trial. If subjects are dissatisfied with the conduct of the trial but have not withdrawn, the investigator should make an effort to address their concerns and retain them in the trial if possible. In doing so, investigators must be careful that the efforts do not cross over into coercion. Investigators should encourage a subject to remain in the study even if the investigational product administration is stopped so that safety information can be collected.

Participation in a clinical trial is voluntary. A subject can withdraw from the study at any time. The sponsor may terminate the study for medical or administrative reasons. An investigator may decline to participate in the conduct of the study if either the investigator or the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) determines that, based on good medical judgment, immediate cessation is appropriate for subject safety. If a decision is made to withdraw a subject from the study, no further investigational product should be administered. Even if the subject discontinues study medication, every attempt should be made to complete all required study evaluations and procedures. Reasons for all withdrawals should be recorded on the CRF. Examples of reasons for withdrawal include:

- 1. A protocol violation has occurred,
- 2. A serious or intolerable adverse event has occurred,
- 3. A clinically significant change in a laboratory parameter has occurred,
- 4. The sponsor or investigator terminates the study, or
- 5. The patient requests to be withdrawn from the study.

Subjects who do not complete the study but who have received investigational product should have a follow-up examination, including a physical examination, vital signs, ECG and clinical laboratory tests according to Section 7.6.

Subjects who withdraw from the study will not be replaced.

## 6.18 Appropriateness of Measurements

The percentage of HbA1c is a widely used measure of chronic glycemia, reflecting average blood glucose levels over a 2- to 3-month period of time. It is an accepted surrogate marker of risk of microvascular complications and is widely used as a measurement for the adequacy of glycemic management. Other study procedures and measurements in this protocol are widely used and generally recognized as reliable, accurate, and relevant for subjects with T2DM.


#### 7 STUDY ACTIVITIES

The study activities at each clinic visit listed below are presented in Appendix 1. The required laboratory tests scheduled at each visit are listed in Appendix 2. Detailed study procedures are described in Section 6.

A visit window of  $\pm$  3 days is allowed for all visits except Visit V6. Visit V6 is the day of randomization and is the basis for all subsequent visit windows.

#### 7.1 Screening Period

7.1.1 Visit V1 (3 days to 3 weeks for metformin-only group and up to 9 weeks for metformin-and-OHA group before run-in period)

The screening can be performed from 3 days to 3 weeks before the start of the wash-out period for subjects who are metformin-and-OHA treated and 3 days to 3 weeks before the start of the run-in period for subjects who are metformin-only treated. At the screening visit, the staff at the investigational site will:

- Explain the content of the informed consent materials to the subject and collect signed informed consent
- Evaluate inclusion and exclusion criteria based on the information collected at the screening visit. Verify compliant fasting status as described in Section 6.9.2.1.
- Obtain medical history and demographic information
- Perform an abbreviated physical examination and record body weight and height
- Measure vital signs, including blood pressures and heart rate
- Perform a 12-lead ECG measurement
- Draw blood if a minimum 10 h fast has been completed by the subject as described in Section 6.9.2.1. The specific laboratory tests scheduled for this visit are listed in Appendix 2.
- Collect a clean-catch, mid-stream urine sample

# 7.2 Wash-out and Run-in Period (Up to 8 weeks prior to randomization)

The wash-out and run-in period is required for any enrolled subject who is taking metformin and one additional OHA. Eligible subjects who are taking metformin only will enter the run-in period directly.

#### 7.2.1 Wash-out Period (Visits V2 and V3)

Two visits will be conducted during the wash-out period. V2 is an on-site clinic visit. At V3 each subject will be evaluated by the investigator or study staff via a phone interview.


#### 7.2.1.1 Visit V2 (8 weeks prior to randomization)

- Evaluate inclusion and exclusion criteria based on the information collected at the screening visit. Verify compliant fasting status as described in Section 6.9.2.1.
- Counsel subject on appropriate diet and exercise (for subjects who are metformin-and-OHA treated)
- Dispense glucometer and instruct subject in SMBG determination and recording (for subjects who are metformin-and-OHA treated)
- Start wash-out and discontinue the non-metformin OHA
- Assess adverse events and potential DKA
- Record pre-treatment medications

#### 7.2.1.2 Visit V3 (6 weeks prior to randomization, off-site phone visit)

- Review SMBG and glycemic control record
- Assess adverse events and potential DKA
- Record pre-treatment medications

#### 7.2.2 Run-in Period

#### 7.2.2.1 Visit V4 (2 weeks prior to randomization)

- Counsel subject on appropriate diet and exercise (for subjects who receive metformin only and do not need a washout)
- Dispense glucometer and instruct subject in SMBG determination and recording (for subjects who receive metformin-only)
- Review SMBG and glycemic control record (for subjects who receive metformin + 1 OHA)
- Dispense run-in kits for run-in period
- Measure vital signs, including blood pressures and heart rate
- Assess adverse events and potential DKA
- Record pre-treatment medications

#### 7.2.2.2 Visit V5 (3 to 5 days prior to randomization)

- Evaluate inclusion and exclusion criteria based on the information collected at the screening visit. Verify compliant fasting status as described in Section 6.9.2.1.
- Perform a complete physical examination and record body weight
- Review SMBG and glycemic control record
- Measure vital signs, including blood pressures and heart rate
- Perform a 12-lead ECG measurement
- Draw blood if a minimum 10 h fast has been completed by the subject as described in Section 6.9.2.1. The specific laboratory tests scheduled for this visit are listed in Appendix 2.
- Collect a clean-catch, mid-stream urine sample
- Assess adverse events and potential DKA
- Record pre-treatment medications


#### 7.3 Treatment Period (Day 1 to Week 96)

At the end of the run-in period, subjects who have successfully completed run-in period and continue to meet the inclusion/exclusion criteria will be randomized and enter the treatment period.

#### 7.3.1 Visit V6 (Day 1 of Week 1)

Visit V6, day of randomization, must be conducted after the HbA1c value from the sample of Visit V5 is available for eligibility confirmation.

- Complete EQ-5D-3L questionnaire
- · Review SMBG and glycemic control record
- Collect used run-in medications and dispense investigational products based on randomization
- Assess adverse events and potential DKA
- Record concomitant medications

#### 7.3.2 Visit V7 (Week 2)

- Review SMBG and glycemic control record
- Measure vital signs, including blood pressures and heart rate
- Collect used study medication, if applicable, and dispense glimepiride based on uptitration criteria assessment
- Assess adverse events and potential DKA
- Record concomitant medications

#### 7.3.3 Visit V8 (Week 4)

- Review SMBG and glycemic control record
- Measure vital signs, including blood pressures and heart rate
- Collect used study medication, if applicable, and dispense glimepiride based on uptitration criteria assessment
- Assess adverse events and potential DKA
- Record concomitant medications

#### 7.3.4 Visit V9 (Week 6)

- Perform an abbreviated physical examination and record body weight
- Review SMBG and glycemic control record
- Measure vital signs, including blood pressures and heart rate
- Collect used study medication, if applicable, and dispense glimepiride based on uptitration criteria assessment
- Draw blood if a minimum 10 h fast has been completed by the subject as described in Section 6.9.2.1. The specific laboratory tests scheduled for this visit are listed in Appendix 2.


- Collect a clean-catch, mid-stream urine sample
- Assess adverse events and potential DKA
- Record concomitant medications

#### 7.3.5 Visit V10 (Week 12)

- Review SMBG and glycemic control record
- Record body weight
- Measure vital signs, including blood pressures and heart rate
- Collect used study medications and dispense investigational products
- Draw blood if a minimum 10 h fast has been completed by the subject as described in Section 6.9.2.1. The specific laboratory tests scheduled for this visit are listed in Appendix 2.
- Collect a clean-catch, mid-stream urine sample
- Assess adverse events and potential DKA
- Record concomitant medications

#### 7.3.6 Visit V11 (Week 24)

- Complete EQ-5D-3L questionnaire
- Perform an abbreviated physical examination and record body weight
- Review SMBG and glycemic control record
- Measure vital signs, including blood pressures and heart rate
- Perform a 12-lead ECG measurement
- Collect used study medications and dispense investigational products
- Draw blood if a minimum 10 h fast has been completed by the subject as described in Section 6.9.2.1. The specific laboratory tests scheduled for this visit are listed in Appendix 2.
- Collect a clean-catch, mid-stream urine sample
- Assess adverse events and potential DKA
- Record concomitant medications

#### 7.3.7 Visit V12 (Week 36)

- Perform an abbreviated physical examination and record body weight
- Review SMBG and glycemic control record
- Measure vital signs, including blood pressures and heart rate
- Collect used study medications and dispense investigational products
- Draw blood if a minimum 10 h fast has been completed by the subject as described in Section 6.9.2.1. The specific laboratory tests scheduled for this visit are listed in Appendix 2.
- Collect a clean-catch, mid-stream urine sample
- Assess adverse events and potential DKA
- Record concomitant medications


#### 7.3.8 Visit V13 (Week 48)

- Perform an abbreviated examination and record body weight
- Review SMBG and glycemic control record
- Measure vital signs, including blood pressures and heart rate
- Collect used study medications and dispense investigational products
- Draw blood if a minimum 10 h fast has been completed by the subject as described in Section 6.9.2.1. The specific laboratory tests scheduled for this visit are listed in Appendix 2.
- Collect a clean-catch, mid-stream urine sample
- Assess adverse events and potential DKA
- Record concomitant medications

#### 7.3.9 Visit V14 (week 60)

- Complete EQ-5D-3L questionnaire
- Perform a complete physical examination and record body weight
- Review SMBG and glycemic control record
- Measure vital signs, including blood pressures and heart rate
- Perform a 12-lead ECG measurement
- Collect used study medications and dispense investigational products
- Draw blood if a minimum 10 h fast has been completed by the subject as described in Section 6.9.2.1. The specific laboratory tests scheduled for this visit are listed in Appendix 2.
- Collect a clean-catch, mid-stream urine sample
- Assess adverse events and potential DKA
- Record concomitant medications

#### 7.3.10 Visit V15 (week 72)

- Perform an abbreviated physical examination and record body weight
- Review SMBG and glycemic control record
- Measure vital signs, including blood pressures and heart rate
- Collect used study medications and dispense investigational products
- Draw blood if a minimum 10 h fast has been completed by the subject as described in Section 6.9.2.1. The specific laboratory tests scheduled for this visit are listed in Appendix 2.
- Collect a clean-catch, mid-stream urine sample
- Assess adverse events and potential DKA
- Record concomitant medications

#### 7.3.11 Visit V16 (week 84, off-site phone visit)

- Review SMBG and glycemic control record
- Assess adverse events and potential DKA
- Record concomitant medications


#### 7.3.12 Visit V17 (end of treatment, week 96)

- Complete EQ-5D-3L questionnaire
- Perform an abbreviated physical examination and record body weight
- Review SMBG and glycemic control record
- Measure vital signs, including blood pressures and heart rate
- Perform a 12-lead ECG measurement
- Draw blood if a minimum 10 h fast has been completed by the subject as described in Section 6.9.2.1. The specific laboratory tests scheduled for this visit are listed in Appendix 2.
- Collect a clean-catch, mid-stream urine sample.
- Collect used investigational products
- Assess adverse events and potential DKA
- Record concomitant medications

### 7.4 Visit V18 (Exit Visit or Early Termination Visit)

- 7.4.1 Visit V18 (week 98 or two weeks after the last dose of investigational product is administered or if a subject withdraws consent)
- Perform a complete physical examination and record body weight
- Review SMBG and glycemic control record
- Measure vital signs, including blood pressures and heart rate
- Draw blood if a minimum 10 h fast has been completed by the subject as described in Section 6.9.2.1. The specific laboratory tests scheduled for this visit are listed in Appendix 2.
- Collect a clean-catch, mid-stream urine sample
- Collect used investigational products if early termination
- Assess adverse events and potential DKA
- Record concomitant medications

## 7.5 Discontinuation of Investigational Product Administration

Subjects who discontinue the investigational product administration early but are willing to remain in the study to allow safety information to be collected should complete the End of Treatment visit procedures. Safety data may be documented following the scheduled clinic visit and/or phone interview procedures as much as possible without the study drug dispensation and accountability procedures. Alternative follow-up methods to allow safety assessment to be recorded may be implemented as unscheduled visits.

## 7.6 Early Termination Procedures

Subjects who withdraw consent and have received investigational products should have a follow-up examination, including a complete physical examination, vital signs, ECG, and


clinical laboratory tests (hematology, serum chemistry, and glycemic control). The sponsor must be notified in the event that a subject withdraws or has been withdrawn from the study.

#### 8 QUALITY CONTROL AND ASSURANCE

The clinical research facility will be monitored by the study monitor to ensure correct performance of the study procedures and to ensure that the study is conducted according to the protocol and relevant regulatory requirements. CRF entries will be verified with the source documentation.

Quality control principles will be applied throughout the performance of this study by following the Standard Operating Procedures (SOPs) of the contract research organization (CRO) and the sponsor. Review procedures will be implemented at the CRO for all documents that are generated in relation to the study.

#### 9 PLANNED STATISTICAL METHODS

#### 9.1 General Considerations

The following sections provide a summary of the planned analysis of the trial but a complete statistical analysis plan will be developed as a separate document and will be the final plan. All statistical analyses will be performed using SAS Version 9.2 or higher.

In general, descriptive statistics (number of subjects [N], mean, standard deviation [SD], Q1, median, Q3, minimum and maximum) will be presented for continuous variables, and frequency and percentage for categorical variables.

The primary efficacy non-inferiority test will be one-sided at 0.025 significance level. The upper bound of the 95% confidence interval (CI) on the difference of HbA1c reduction between bexagliflozin and glimepiride will be used to determine the study's conclusion. That is, if the upper bound of the CI is within 0.35%, then the primary objective of the study is met. Superiority will be declared without additional statistical testing when the upper bound of the 95% CI for the difference in change from baseline at week 60 in HbA1c comparing bexagliflozin group with glimepiride group is less than 0.

The secondary efficacy objectives will be tested at two-sided 0.05 significance level following a sequential testing procedure to control the overall type I error of 0.05. The secondary efficacy endpoints will be tested only if the primary efficacy assessment achieves significance, and following the hierarchy as below:

- 1. Superiority test of the change in body weight in subjects with baseline BMI  $\geq$  25 kg/m<sup>2</sup> in the bexagliflozin group compared with glimepiride group at week 60
- 2. Superiority test of the change in SBP in subjects with baseline SBP ≥140 mmHg in the bexagliflozin group compared with glimepiride group at week 60
- 3. Superiority test of the difference in proportion of subjects with ≥1 severe or documented symptomatic hypoglycemia events in the bexagliflozin group compared with glimepiride group over 96 weeks

The exploratory efficacy objectives and safety objectives will be analyzed descriptively.

## 9.2 Determination of Sample Size

Approximate total 420 subjects will be randomized and equally allocated to receive bexagliflozin tablets 20 mg or placebo, and glimepiride capsules, 2 mg, 4 mg, 6 mg or placebo.

The sample size calculation for this study is based on a two group t-test with a one-sided significance at the 0.025 level and the following assumptions:

1. The non-inferiority limit (margin) for mean change from baseline to week 60 in HbA1c comparing bexagliflozin group to glimepiride group will be 0.35%


2. The pooled standard deviation for the change from baseline to week 60 in HbA1c for bexagliflozin group and glimepiride group will be 1.0%

Theracos Sub, LLC

27 October 2016

Under the above assumptions, an estimated sample size of 172 patients is needed in each treatment arm to detect non-inferiority of bexagliflozin to glimepiride with respect to change in HbA1c at week 60 from baseline. This estimation is based on a one-sided t-test with 90% power at a 0.025 level of significance. A sample size of 210 per arm has been selected to account for approximate 18% drop-out rate and to allow adequate safety evaluation. The total sample size for this study will be 420 subjects.

This study will be conducted at multiple investigative sites and will likely involve various numbers of subjects at each site. Enrollment will be on a competitive basis, but will be capped at 40 subjects from each site.

#### 9.3 Analysis Populations

#### 9.3.1 Intention-to-Treat Analysis set

All subjects who are randomized regardless of treatment adherence or availability of follow-up data will be included in the intention-to-treat analysis set (ITT). All analyses of the ITT will be based on each subject's randomized assigned treatment. The ITT analysis set will serve as the primary set for the efficacy analyses.

#### 9.3.2 Safety Analysis Set

All subjects who are randomized and take at least one dose of double-blind study medication will be included in the Safety Analysis Set. Safety analyses will be based on the medication that was actually taken by each subject. The Safety Analysis Set is the primary analysis set for safety evaluation.

#### 9.3.3 Per Protocol Analysis Set

The Per Protocol (PP) Analysis Set will include all subjects in the ITT who meet the study eligibility requirements and have no major protocol deviations that affect the validity of the efficacy measurements. Protocol deviations that may result in subject exclusion from the PP Analysis Set will be detailed in the Statistical Analysis Plan. The subject assignment to the PP analysis set will be determined prior to database lock. The PP analysis set will serve as the secondary set for efficacy assessments.

## 9.4 Demographics and Baseline Characteristics

Demographic and baseline characteristics will be summarized descriptively based on the ITT and PP analysis set for each treatment group as well as for all subjects combined. Key variables include age, gender, race, ethnicity, baseline HbA1c values, blood pressure, body weight, body mass index (BMI in kg/m²), fasting plasma glucose level, eGFR, duration of diabetes and prior anti-diabetic treatment status at screening (including type of therapy used [metformin, sulfonylurea, DPP-4 inhibitor, alpha-glucosidase inhibitor etc.]). In general,


baseline measurement is defined as the last measurement prior to the first dose of doubleblind medication.

#### 9.4.1 Concomitant Medications

Concomitant medications will be coded using the World Health Organization Drug Dictionary (WHO-DD), and include medications that are either started prior to the study treatment and continue to be taken during the study treatment period, or medications started after the start of study treatment. Concomitant medications will be summarized by ATC term and by treatment groups.

#### 9.5 Primary Efficacy Analyses

#### 9.5.1 Hypotheses for the Primary Endpoint

The null and alternative hypotheses for the primary endpoint are:

H<sub>0</sub>: 
$$\mu$$
 bexagliflozin -  $\mu$  comparator  $\geq \delta$   
H<sub>a</sub>:  $\mu$  bexagliflozin -  $\mu$  comparator  $\leq \delta$ 

Where  $\mu_{bexagliflozin}$  and  $\mu_{comparator}$  represent the mean change in HbA1c at week 60 from baseline for bexagliflozin and comparator groups, respectively. Non-inferiority margin  $\delta$  is chosen to be 0.35% using clinical judgment, with reference to relevant regulatory guidance.

#### 9.5.2 Statistical Methods for Primary Analyses

For the primary endpoint, the treatment difference will be examined by using a mixed model repeated measures (MMRM) analysis of covariance model (ANCOVA). The model will include treatment, visit, treatment-by-visit interaction and randomization stratification factors as the fixed effects terms and the baseline HbA1c value as a fixed effect covariate. Least squares mean treatment differences between the bexagliflozin group and the comparator group at week 60 will be estimated from the model. An unstructured covariance will be used to model the within-subject correlation. If the model with the unstructured covariance structure does not converge, an autoregressive(1) covariance structure will be used.

HbA1c values obtained after the start of rescue medication will not be excluded in the analysis. These analyses will be conducted on both ITT (primary) and PP analysis sets, and conclusions can be considered more robust when both approaches support the non-inferiority of the treatment.

In non-inferiority analysis, a CI is calculated to estimate the range of values in which the treatment difference is likely to lie. This CI is used to provide the basis for drawing the study's conclusions. In this specific test, if the 95% CI lies below the specified non-inferiority margin 0.35%, the results would lead to a conclusion of non-inferiority of bexagliflozin treatment to glimepiride treatment. Superiority of bexagliflozin group over


glimepiride group at week 60 in HbA1c change from baseline will be declared if the upper bound of 95% CI is less than 0.

Sensitivity analyses will also be performed as the following, and these analyses will be conducted for ITT and PP analysis sets.

- 1. Missing data will be imputed via multiple imputations, following which the MMRM will be repeated on the complete datasets with results combined across complete datasets using standard MI techniques; HbA1c values collected after the start of rescue medication will not be excluded.
- 2. Missing data will be imputed via LOCF, following which the MMRM will be repeated; HbA1c values collected after the start of rescue medication will be considered missing.
- 3. HbA1c values collected after the start of rescue medication will be considered missing, and the MMRM analyses will be re-performed.

#### 9.5.3 Analysis of Dropouts Pattern

The early termination rate is estimated to be 18%. To the extent possible, attempts will be made to minimize the amount of missing data through measures planned in the study conduct.

The number, timing, pattern, reason for and possible implications of missing values in efficacy assessments will be investigated. The dropout patterns will be assessed by Kaplan-Meier plots if applicable to assess whether they differ between treatment groups.

## 9.6 Secondary Efficacy Analyses

To assess the treatment effect on the change of body weight in subjects with baseline BMI  $\geq$  25 kg/m² at week 60, an analysis of covariance model (ANCOVA) will be implemented using all available data at week 60 (values obtained after the start of rescue medication will not be excluded in the analysis). The model will include treatment, randomization stratification factors, and the baseline weight value as fixed effects/covariates. Least squares mean treatment differences between the bexagliflozin group and the comparator group will be estimated from the model. The corresponding 95% CI and p-value will be provided.

The change in systolic blood pressure (SBP) in subjects with baseline SBP  $\geq$  140 mmHg in the bexagliflozin group compared with glimepiride group at week 60 will be analyzed using the same method.

The difference in proportion of subjects with  $\geq 1$  severe or documented symptomatic hypoglycemia events in the bexagliflozin group compared with glimepiride group over 96 weeks will be analyzed using logistic regression model which includes terms of treatment, randomization stratification. Odd ratio estimates, 95% two-sided confidence intervals and p-values for the treatment difference will be provided.


All analyses will be conducted in ITT analysis set. A hierarchical testing procedure will be applied to above three endpoints in the sequence provided above.

#### 9.7 Other Efficacy Analyses

Changes in FPG, SBP/DBP, and body weight for all subjects during the treatment period will be summarized descriptively by each time point (i.e., Weeks 2, 4, 6, 12, 24, ..., etc.). In addition, these endpoints may be analyzed using a similar MMRM model as used for the primary analysis of HbA1c to compare two treatment groups.

Cumulative summary on the proportion of subjects achieving HbA1c < 7%, and the proportion of subjects with documented hypoglycemia event will be presented over time. Generalized estimation equation (GEE) method may be utilized for assessment of treatment effects.

Analyses will be conducted using ITT analysis set.

#### 9.8 Analysis of Safety

Safety data include AEs, physical exam results, vital signs, ECG results, and clinical lab results including serum chemistry, hematology, serum lipids, glycemic control parameters and urinalysis. Observed data will be summarized by treatment using safety analysis set.

#### 9.8.1 Adverse Events

AEs will be mapped to preferred term and body system using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary. AEs that begin at or after the first administration of double-blind study medication or existing AEs that worsen in severity after the first dose of double-blind study medication are considered treatment emergent AEs (TEAE). The number and percentage of subjects reporting TEAEs will be summarized for each treatment group by MedDRA system organ class and preferred term. Further summaries by severity, and by relationship to study treatment will also be provided. Drug-related adverse events will be considered those to be at least possibly related to the study treatments based on the investigators assessment.

The number and percentage of subjects reporting serious AEs, and the number and percentage of subjects reporting AEs leading to treatment discontinuation will also be summarized for each treatment group by MedDRA system organ class and preferred term.

#### 9.8.2 Adverse Events of Special Interest

AE of special interest include UTI, GMI, diuretic effects, hepatotoxicity, cardiovascular events, hypoglycemia, fracture, malignancy, hypersensitivity reactions, hypotensive episodes, DKA, renal failure events, and amputation. These AEs of special interest will be prospectively identified based on the MedDRA preferred terms in the adverse event log by a medical expert prior to the data base lock and unblinding of the individual subject treatment assignment. The list of adverse events of special interest will be confirmed in a peer review process.


The number and percentage of subjects experienced TEAE of special interest will be summarized for each treatment group by types of events. The incidence rate of adverse events of special interest per 100 patient years will also be summarized. Additional analyses will be specified in the statistical analysis plan to evaluate other event associated safety parameters and potential risks in subpopulations based on age, gender, or other baseline characteristics.

#### 9.8.3 Clinical and Laboratory Events and Analyses

Clinical laboratory (see Section 6 for a complete list), vital signs, and 12-lead ECG will be measured at scheduled visits (see Appendix 1). These data will be summarized as actual values and changes from baseline by treatment for each visit for selected parameters.

Laboratory data will be classified as low, normal or high relative to the parameter's reference range. Laboratory abnormalities for each treatment will also be summarized with shift tables for selected parameters.

#### 9.8.4 Physical Examination

Physical examination findings will be presented in a by subject listing.

#### 9.9 Health Related Quality of Life Assessment

Descriptive statistics will be calculated for each item of the questionnaire, the EQ-5D-3L index score and visual analog score. Both actual values and changes from baseline will be summarized by treatment group for each visit. In addition, the changes from baseline in index score and visual analog score will be assessed for treatment effect using MMRM method. Similar to efficacy endpoints, the model will include treatment, visit, treatment-by-visit interaction and randomization stratification factors as the fixed effects terms and the baseline EQ-5D-3L index score (or visual analog score) as a fixed effect covariate.

#### 9.10 Interim Analysis

No interim analysis will be performed during this study.

## 9.11 Final Analysis

After all subjects have completed the planned 60 weeks of blinded study treatment and the subsequent safety extension and follow-up periods, the final analysis of the clinical study will be completed. At this time, the database will be cleaned and locked, and the treatment codes will be unblinded.


#### 10 ADMINISTRATIVE CONSIDERATIONS

#### 10.1 Investigators and Study Administrative Structure

Information regarding key personnel involved in the conduct of the study, including names and contact details of participating investigators, monitors, clinical laboratories, and technical departments and/or institutions, as well as information on members of additional study committees, will be found in the study files of the investigational site.

## 10.2 Institutional Review Board (IRB) or Independent Ethics Committee (IEC) Approval

The study protocol, informed consent document, relevant supporting information, and all types of subject recruitment or advertisement information must be submitted to the IRB/IEC for review and must be approved by the sponsor and the IRB/IEC before the study is initiated. Any amendments or addenda to the protocol must also be approved by the IRB/IEC prior to implementing changes in the study. The investigator is responsible for keeping the IRB/IEC informed of the progress of the study and of any changes made to the protocol as deemed appropriate, but in any case at least once a year. The investigator must also keep the IRB/IEC informed of any SAEs occurring to subjects under their supervision.

#### 10.3 Ethical Conduct of the Study

The procedures set out in this protocol pertaining to the conduct, evaluation, and documentation of this study are designed to ensure that the sponsor and investigator follow ICH Good Clinical Practice (GCP) Guidelines and the guiding principles detailed in the Declaration of Helsinki. The study will also be carried out in keeping with applicable local laws and regulations. An inspection by the sponsor representatives and/or their designee and/or other authorized regulatory authorities representatives may occur at any time. The investigator must agree to the inspection of study-related records by the regulatory authority/sponsor representatives, and must allow direct access to source documents to the regulatory authority/sponsor representatives.

The investigator is responsible for complying with the protocol and all appropriate regulations and guidelines governing global clinical research. Additionally, he/she is responsible for ensuring that all participating staff members are adequately trained and competent to perform his/her assigned tasks.

Modifications to the study protocol will not be implemented by either the sponsor or the investigator without agreement by both parties. However, the investigator may implement a deviation from or a change of the protocol to eliminate any immediate hazards to the trial subjects without prior IRB/IEC or sponsor approval/favorable opinion. As soon as possible, the implemented deviation or change, the reasons for it, and if appropriate, the proposed protocol amendment should be submitted to the IRB/IEC and sponsor.


Any deviations from the protocol must be fully explained and documented by the investigator. The circumstances, action taken, and impact of the deviation on the trial must be communicated by the principal investigator to the designated medical monitor. Any subsequent actions will be assessed by the designated medical monitor and documented.

#### 10.4 Subject Information and Consent

Prior to the beginning of the study, the investigator must have received from the IEC or IRB the written approval or favorable opinion of the informed-consent form and any other written information to be provided to subjects. The written approval of the IRB/IEC together with the approved subject information/ informed consent forms must be filed. The informed consent form must contain all elements required by authorized regulatory authorities and the ICH GCP guidelines (E6), in addition to, any other elements required by local regulations or institutional policy.

Written informed consent must be obtained before any study-specific procedure takes place. Participation in the study and date of informed consent given by the subject should be documented appropriately in the subject's files. A copy of the signed informed consent form must be provided to the subject. If applicable, it will be provided in a certified translation in the language understood by the subject, if not English. Signed consent forms must remain in each subject's study file and must be available for verification by study monitors at any time.

#### 10.5 Subject Confidentiality

The information obtained during the conduct of this clinical study is confidential, and disclosure to third parties other than those noted below is prohibited. Information obtained during the conduct of this study will be used by the sponsor in connection with the development of the investigational product. The study investigator is obliged to provide the sponsor with complete test results and all data developed in this study. Subject-specific information may be provided to other appropriate medical personnel only with the subject's permission. To ensure compliance with current ICH guidelines, data generated by this study must be available for inspection upon request by representatives of national and local health authorities, the sponsor, and the IRB/IEC for each study site. Study information from this protocol will be posted on clinicaltrials.gov and any local regulatory registry websites, as required by regulation.

Subject names and other identifiers, such as photographs, audio, or videotapes, may not be disclosed in any publication without prior written authorization from the subject.

## 10.6 Study Monitoring

An authorized sponsor representative will conduct site visits to inspect study data, subjects' medical records, and CRFs in accordance with ICH guidelines, GCPs, and the respective national and local government regulations and guidelines.


The investigator will permit authorized representatives of the sponsor and the respective national or local health authorities, other authorized regulatory authorities, and IRB/IEC to inspect facilities and records relevant to this study.

#### 10.7 Case Report Forms and Study Records

For each subject consented, a case report form (CRF), in paper or electronic format, will be supplied and maintained by the CRO staff and signed by the investigator or authorized designee to indicate that he/she has reviewed and agrees with the entered data. This also applies to those subjects who fail to complete the trial. The reason a subject is withdrawn must be recorded in the case report form.

Entries made in the CRF must be verifiable against source documents. Source documents are defined as all medical records, medical notes, laboratory results, ECG traces and any additional document other than the CRF that has original subject information contained within it.

All CRFs and source documents should be completed following GCP and the Sponsor or its designees standard operating procedures.

#### 10.8 Data Monitoring Committee

An independent Data and Safety Monitoring Board (DSMB) will monitor overall safety information during the bexagliflozin development program. The safety review activity and potential risk benefit assessments utilized by the DSMB will be defined in its charter.

#### 10.9 Protocol Violations/Deviations

Protocol violations include deviations from the inclusion and exclusion criteria, concomitant medication restrictions, and any other protocol requirement that results in a significant added risk to the patient or has an impact on the quality of the data collected or the outcome of the study. A deviation occurs when there is non-adherence to study procedures or schedules, as specified by the protocol, which does not involve inclusion/exclusion criteria or the primary endpoint and which does not place the patient at any added risk or affect the data quality or study outcome. Examples of deviations may include common out-of-window visits, a missed procedure, etc. Protocol violations will reported in the final clinical study report, whereas protocol deviations may be mentioned but are not required to be reported.

It is important to conduct the study according to the protocol. Protocol deviation waivers will not be prospectively granted by the sponsor. If minor protocol deviations occur, the investigator must decide the most appropriate way to proceed with study activities and should consult the study representative for assistance. If major protocol deviations occur, the sponsor's Medical Monitor must be notified immediately so that a decision about whether to keep the subject in the study can be made.

Only when an emergency occurs that requires a departure from the protocol for an individual subject can there be a departure without the sponsor's pre-approval. The nature and reasons


for the protocol deviation/violations will be recorded in the subject's CRF, and the principal investigator must notify the sponsor.

Protocol deviations/violations must be reported in the final study report.

#### 10.10 Access to Source Documentation

Authorized sponsor representatives will conduct site visits to inspect study data, subjects' medical records, and CRFs in accordance with ICH guidelines, GCPs, and the respective local and national government regulations and guidelines.

The investigator will permit authorized representatives of the sponsor and the respective national or local health authorities, other authorized regulatory authorities, and IRB/IEC to inspect facilities and records relevant to this study.

Each center will be visited at regular intervals by a monitor to ensure compliance with the study protocol, GCP, and legal aspects. This will include on-site checking of the CRFs for completeness and clarity, cross-checking with source documents, and clarification of administrative matters.

All CRF data will be entered into a clinical database. Following the correction of any errors, the clinical database will be locked.

#### 10.11 Retention of Data

The study file and all source data should be retained until notification is given by the sponsor for destruction.

If the investigator withdraws from the trial and relinquishes his/her responsibility for the maintenance and retention of records, he/she must notify the sponsor in writing so that arrangements can be made to properly store the trial materials.

## 10.12 Publication and Disclosure Policy

All data and results and all intellectual property rights in the data and results derived from the study will be the property of the sponsor, who may utilize the data in various ways, such as for submission to government regulatory authorities or disclosure to other investigators.

No publication or disclosure of study results will be permitted except as specified in a separate, written agreement between Theracos Sub LLC and the investigator. If results of this study are reported in medical journals or at meetings, all subjects' identities will remain confidential.


#### 11 REFERENCE LIST

IDF (2015). "International Diabetes Federation Diabetes Atlas Seventh Edition."

Look, A. R. G., R. R. Wing, et al. (2013). "Cardiovascular effects of intensive lifestyle intervention in type 2 diabetes." N Engl J Med 369(2): 145-154.

Nauck, M. A. (2014). "Update on developments with SGLT2 inhibitors in the management of type 2 diabetes." Drug Design, Development and Therapy 8: 1335-1380.

Santer, R., M. Kinner, et al. (2003). "Molecular analysis of the SGLT2 gene in patients with renal glucosuria." J Am Soc Nephrol 14(11): 2873-2882.

Scheen, A. J. and L. F. Van Gaal (2014). "Combating the dual burden: therapeutic targeting of common pathways in obesity and type 2 diabetes." Lancet Diabetes Endocrinol 2(11): 911-922.

Schwartz, S., A. N. Fabricatore, et al. (2012). "Weight reduction in diabetes." Adv Exp Med Biol 771: 438-458.

Seufert, J. (2015). "SGLT2 inhibitors - an insulin-independent therapeutic approach for treatment of type 2 diabetes: focus on canagliflozin." Diabetes Metab Syndr Obes 8: 543-554.

Van den Heuvel, L. P., K. Assink, et al. (2002). "Autosomal recessive renal glucosuria attributable to a mutation in the sodium glucose cotransporter (SGLT2)." Hum Genet 111(6): 544-547.

Zhang, W., A. Welihinda, et al. (2011). "EGT1442, a potent and selective SGLT2 inhibitor, attenuates blood glucose and HbA(1c) levels in db/db mice and prolongs the survival of stroke-prone rats." Pharmacol Res 63(4): 284-293.


## Appendix 1 Schedule of Events

| | Screening | Wasi | h-out | Ru | n-in | | | | Effica | cy Asse | ssment | | | | Safe | ty Exte | nsion | Follow-<br>up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit number | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12 | V13 | V14 | V15 | V16 | V17 | V18 |
| Time to Randomization Visit (wk) | -11 | -8 | -6 | -2 | -0.5 | 0 | 2 | 4 | 6 | 12 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | 98 |
| Off-site phone visit | | | X | | | | | | | | | | | | | X | | |
| Informed Consent | X | | | | | | | | | | | | | | | | | |
| EQ-5D-3L | | | | | | X | | | | | X | | | X | | | X | |
| Screening for I/E criteria | X | X | | | X | | | | | | | | | | | | | |
| Demographics and medical history | X | | | | | | | | | | | | | | | | | |
| Diet & exercise counseling | | X | | X | | | | | | | | | | | | | | |
| Physical exam | | | | | X | | | | | | | | | X | | | | X |
| Abbreviated physical exam | X | | | | | | | | X | | X | X | X | | X | | X | |
| Record height | X | | | | | | | | | | | | | | | | | |
| Record body weight | X | | | | X | | | | X | X | X | X | X | X | X | | X | X |
| Dispense diary & glucometer | | X | | X | | | | | | | | | | | | | | |
| Diary & glucometer record review | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Start wash-out | | X | | | | | | | | | | | | | | | | |
| Dispense Run-in Medication | | | | X | | | | | | | | | | | | | | |
| Randomization | | | | | | X | | | | | | | | | | | | |
| Vital signs | X | | | X | X | | X | X | X | X | X | X | X | X | X | | X | X |
| ECG | X | | | | X | | | | | | X | | | X | | | X | |
| Discontinue non-metformin OHA | | X | | | | | | | | | | | | | | | | |
| Dispense bexagliflozin | | | | | | X | | | | X | X | X | X | X | X | | | |
| Dispense glimepiride | | | | | | X | X | X | X | X | X | X | X | X | X | | | |
| Blood draw for clinical lab test | X | | | | X | | | | X | X | X | X | X | X | X | | X | X |
| Urine collection | X | | | | X | | | | X | X | X | X | X | X | X | | X | X |
| AE | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Con Med | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

## Appendix 2 Schedule of Clinical Laboratory Tests

| | Screening | Was | h-out | Ru | n-in | | | | Eff | icacy A | ssessm | ent | | | Safe | y Exte | nsion | Follow-<br>up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12 | V13 | V14 | V15 | V16 | V17 | V18 |
| Time to Randomization Visit (weeks) | -11 | -8 | -6 | -2 | -0.5 | 0 | 2 | 4 | 6 | 12 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | 98 |
| Hematology | X | | | | X | | | | X | | X | | X | X | | | X | X |
| Serum chemistry electrolytes | X | | | | X | | | | X | | X | | X | X | | | X | X |
| Fasting Plasma Glucose | X | | | | X | | | | X | X | X | X | X | X | X | | X | X |
| HbA1c | X | | | | X | | | | | X | X | X | X | X | X | | X | X |
| Lipids | X | | | | X | | | | | | X | | | X | | | X | X |
| Urinalysis | X | | | | X | | | | X | X | X | X | X | X | X | | X | X |
| Urine pregnancy test (UPT) | X | | | | X | | | | X | X | X | X | X | X | X | | X | X |

## Appendix 3 Sponsor Signatures

Study Title:

A Phase 3, Randomized, Double-Blind, Active-Controlled Study to

Evaluate the Effects of Bexagliflozin versus Glimepiride in Subjects with Type 2 Diabetes Mellitus Who Have Inadequate Glycemic

Control by Metformin

Study Number:

THR-1442-C-480

V 3.0 Final Date:

27 October 2016

This clinical study protocol was subject to critical review and has been approved by the sponsor. The following personnel contributed to writing and/or approving this protocol:

| - | | | | | - |
|-----|---|----|---|---|---|
| C, | 1 | OT | 3 | 0 | N |
| . 7 | | 20 | ш | | |

Annie Conery, Ph.D.

Protocol Originator

Massachusetts General Hospital Consultant for Theracos Sub, LLC Date:\_\_/0/27/16

Signed:

J. Paul Lock, M.D.

Medical Monitor

Consultant for Theracos Sub, LLC

Signed:

Wenjiong Zhou, Ph.D.

Statistician FMD K&L

Consultant for Theracos Sub, LLC

Date: 270ct 2016

Date:

| Appendix 3 | Sponsor Signatures |
|---|---|
| Study Title: | A Phase 3, Randomized, Double-Blind, Active-Controlled Study to<br>Evaluate the Effects of Bexagliflozin versus Glimepiride in Subjects<br>with Type 2 Diabetes Mellitus Who Have Inadequate Glycemic<br>Control by Metformin |
| Study Number: | THR-1442-C-480 |
| V 3.0 Final Date: | 27 October 2016 |
| Signed: Annie Conery Protocol Origi Massachusetts | |
| Signed: J. Paul Lock, Medical Moni Consultant for | |

Signed:

Wenjiong Zhou, Ph.D.

Consultant for Theracos Sub, LLC

Statistician FMD K&L

Date:

Bexagliflozin Tablets Theracos Sub, LLC Clinical Trial Protocol: THR-1442-C-480 27 October 2016

Appendix 4 Investigator's Signature

**Study Title:** A Phase 3, Randomized, Double-Blind, Active-Controlled Study to

Evaluate the Effects of Bexagliflozin versus Glimepiride in Subjects with Type 2 Diabetes Mellitus Who Have Inadequate Glycemic

Control by Metformin

**Study Number:** THR-1442-C-480 **V3.0 Final Date:** 27 October 2016

I have read the protocol described above. I agree to comply with the International Conference on Harmonisation (ICH) Tripartite guideline on Good Clinical Practice (GCP) and all applicable regulations and to conduct the study as described in the protocol.

I agree to ensure that Financial Disclosure Statements will be completed by myself and my subinvestigators at the start of the study and for up to 1 year after the study is completed, if there are changes that affect my financial disclosure status.

I agree to ensure that the confidential information contained in this document will not be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Theracos Sub, LLC.

| Signed: | Date: |
|-----------------------|-------|
| Clinical Investigator | |